# ILLINOIS

### Office of the Vice Chancellor for Research & Innovation

Office for the Protection of Research Subjects 1901 S. First St., Suite A, MC-685 Champaign, IL 61820

## **Notice of Approval: Amendment 10**

September 4, 2023

Principal Investigator Wendy Rogers

CC Raksha Mudar, Elizabeth Lydon, George Mois
Protocol Title Video Technology-based Social Engagement

Protocol Number 22212

Funding Source NIH (2 R44 AG059450-02A1)

**Review Type** Expedited 6, 7

Amendment Requested Research team update

Status Active

**Risk Determination** No more than minimal risk

Amendment Approval Date September 4, 2023 Expiration Date September 14, 2026

This letter authorizes the use of human subjects in the above protocol. The University of Illinois at Urbana-Champaign Institutional Review Board (IRB) has reviewed and approved the research study as described.

The Principal Investigator of this study is responsible for:

- Conducting research in a manner consistent with the requirements of the University and federal regulations found at 45 CFR 46.
- Using the approved consent documents, with the footer, from this approved package.
- Requesting approval from the IRB prior to implementing modifications.
- Notifying OPRS of any problems involving human subjects, including unanticipated events, participant complaints, or protocol deviations.
- Notifying OPRS of the completion of the study.



IRB Number: 22212

## **Human Subjects Research – Protocol Form**

## **Guidelines for completing this research protocol:**

- Please submit typed applications via email. Handwritten forms and hard copy forms will not be accepted.
- For items and questions that do not apply to the research, indicate as "not applicable."
- Provide information for all other items clearly and avoid using discipline specific jargon.
- Please only include text in the provided boxes. The text boxes will expand as they are typed in to accommodate large amounts of text.

## Before submitting this application, ensure that the following have been completed.

- Protocol Form is complete.
- Relevant CITI modules have been completed for all members of the research team at www.citiprogram.org.
- Informed consent/assent/parental permission document(s) are provided.
- Relevant waivers and appendices are provided.
- Recruitment materials are provided.
- Research materials (e.g. surveys, interview guides, etc.) are provided.
- Any relevant letters of support are provided.

Instructions on the non-exempt review process and guidance to submitting applications, can be found on the OPRS <u>website</u>. You may also contact OPRS by email at <u>irb@illinois.edu</u> or phone at 217-333-2670.

**Submit completed applications via email to:** irb@illinois.edu.



## **Section 1: PRINCIPAL INVESTIGATOR (PI)**

| The Illinois <u>Campus Administrative Manual</u> allows assistant, associate, and full professors to act as PI. Other individuals may serve as PI after obtaining approval from the necessary party. | | | |
|---|---|---|---|
| Last Name: Rogers | First Name: Wendy Degree(s): PhD | | |
| Dept. or Unit: Department of Kinesiology and Community Health | Office Address: 3011A | | |
| Street Address: 1206 South Fourth | City: Champaign State: IL Zip Code: 61820 | | |
| Phone: 217-300-1470 | E-mail: wendyr@illinois.edu | | |
| Urbana-Champaign Campus Status: Non-visiting member of (Mark One) Faculty Academic Professional/Staff (Student Investigators cannot serve as PI) | | | |
| Training Required CITI Training, Date of Co Additional training, Date of Complete | | years), Novem | ber 9, 2019 |
| Section 2. RESEARCH TEAM | | | |
| 2A. Are there other investigators eng Yes (include a Research Team Form | _ | | |
| No | | | |
| 2B. If yes, are any of the researchers not affiliated with Illinois? Yes | | | |
| □ No | | | |
| Section 3. PROTOCOL TITLE | | | |
| Video Technology-based Social Engage | ement | | |
| Section 4. FUNDING SOURCE | | | |
| 4A. Is the research funded? | | | |
| Research is <b>not funded</b> and is <b>not pending</b> a funding decision (Proceed to Section 5). | | | |
| Research is <b>funded</b> (funding decision has been made). | | | |
| Funding decision is <b>pending</b> . Funding proposal submission date: 4B. Indicate the source of the funding. | | | |
| University of Illinois Department, ( | | fy: | |
| Federal, please specify: National Ir | | <u>, </u> | |



## **Protocol Form**

| State of Illinois Department or Agency, please specify: Other, please specify: |
|---|
| 4C. Sponsor-assigned grant number, if known: 2 R44 AG059450-02A1 |
| 4D. A complete copy of the funding proposal or contract is attached. |
| Attached, please specify title: Enhancing Quality of Life for Older Adults With and Without MCI |
| through Social Engagement Over Video Technology |
| 4E. Funding Agency Official To Be Notified of IRB Approval (if Applicable) |
| Name: |
| Agency: |
| E-mail: |
| Phone: |
| Section 5. CONFLICTS OF INTEREST |
| Please indicate below whether any investigators or members of their immediate families have any of |
| the following. If the answer to any of the following items is yes, please submit the University of Illinois |
| approved conflict management plan. If you have any questions about conflicts of interest, contact |
| coi@illinois.edu. |
| <b>5A.</b> Financial interest or fiduciary relationship with the research sponsor (e.g. investigator is a consultant |
| for the research sponsor). Yes No |
| <b>5B.</b> Financial interest or fiduciary relationship that is related to the research (e.g. investigator owns a |
| startup company, and the intellectual property developed in this protocol may be useful to the |
| company). 🗌 Yes 🔀 No |
| <u>5C.</u> Two or more members of the same family are acting as research team members on this protocol. |
| Yes No |

### Section 6. SUMMARY & PURPOSE OF RESEARCH

6A. In lay language, summarize the objective and significance of the research.

The goal of this project is to test the efficacy of a social engagement intervention delivered using a video-technology called OneClick for older adults with and without mild cognitive impairment (MCI). Following the baseline assessment, participants will be randomized into two groups: Group 1 (intervention first), or Group 2 (intervention later). Group 1 will receive 8 weeks of the OneClick social engagement intervention, during which time Group 2 will receive no planned intervention. Both groups will receive an assessment at 4 weeks and another assessment at 8 weeks after they are enrolled in the study. Group 2 will then be rolled into the OneClick social engagement intervention. They will receive 8 weeks of the OneClick social

<sup>&</sup>lt;sup>2</sup> Clarify whether or not the sponsor requires the protocol adhere to ICH GCP (E6) standards

| OFFICE FOR THE PROTECTION OF RESEAR | CH SUBJECTS | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | CHAMPAIGN |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 02/07/2020 |

<sup>&</sup>lt;sup>1</sup> Clarify whether or not sponsor requires specific language in the contractual agreement that impacts human subjects research



engagement intervention, similar to Group 1, and will be assessed after four weeks and 8 weeks of participating in the video chat intervention. We will test the benefits of using OneClick over 8 weeks by measuring social engagement, quality of life, and user acceptance of technology.

Older adults are at risk of social isolation, and therefore, negative health and quality-of-life outcomes. For individuals with MCI, social activities and engagement may slow disease progression and the transition into dementia. Social engagement technologies offer a novel opportunity to connect people to enhance social interactions. OneClick's existing platform connects people from across the country and world over shared interests in live, small group video conversations. In distinct contrast to existing social media and online chat, dating, or meet-up platforms, OneClick connects people virtually without the need to exchange private information or download an application. Users of different ages, including older adults, have reported positive experiences using OneClick. Our prior feasibility and usability studies have shown that older adults with and without MCI are interested in and will use computer technology and the internet for personal enjoyment. In an initial project funded by a SBIR Phase I (R43AG069450) grant from NIA, we optimized the OneClick platform for use by older adults with and without MCI (Protocol #18585 and #19145) and completed an experiential field trial to assess usability (Protocol #19271). The current project, funded by a SBIR Phase II grant (2 R44 AG059450-02A1), will test the efficacy of the OneClick social engagement intervention in a larger randomized control trial (RCT) using a wait-list control group design.

| randomized control trial (RCT) using a wait-list control group design. |
|---|
| 6B. Indicate if your research includes any of the following: |
| Secondary data (use of data collected for purposes other than the current research project) |
| Data collected internationally (include <u>International Research Form</u> ) |
| Translated documents (include <u>Certificate of Translation Form</u> and translated documents) |
| Research activities will take place at Carle (include documentation (email or letter) from Carle stating |
| that the review of your Research Services Request Form is complete) |
| 6C. Letters of support from outside institutions or entities that are allowing recruitment, research, or |
| record access at their site(s) are attached. X Yes Not Applicable |
| Section 7. PROCEDURES |
| Section 7. PROCEDURES |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. Surveys or questionnaires, select all that apply: Paper Telephone Online |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. Surveys or questionnaires, select all that apply: Paper Telephone Online Interviews |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. Surveys or questionnaires, select all that apply: Paper Telephone Online Interviews Focus groups |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. Surveys or questionnaires, select all that apply: □ Paper ☑ Telephone ☑ Online Interviews □ Focus groups □ Field work or ethnography |
| Section 7. PROCEDURES 7A. Select all research methods and/or data sources that apply. Surveys or questionnaires, select all that apply: Paper Telephone Online Interviews Focus groups Field work or ethnography Standardized written, oral, or visual tests |



| Intervention or experimental manipulation |
|---|
| Exercise and muscular strength testing |
| Noninvasive procedures to collect biological specimens (e.g., hair and nail clippings, saliva, etc.) |
| Noninvasive procedures to collect physiological data (e.g., physical sensors, electrocardiography, etc.) |
| Procedures involving radiation |
| Recording audio and/or video and/or taking photographs |
| Recording other imaging |
| Materials that have already been collected or already exist, specify source of data: |
| HIPAA-protected data |
| FERPA-protected data |
| GDPR-protected data |
| Other, please specify: |
| 7B. List all testing instruments, surveys, interview guides, etc. that will be used in this research. |
| Telephone screening DRAFT |
| Modified Telephone Interview for Cognitive Status (TICS-M) |
| Modified Techsage Background Questionnaire (TBSQ) |
| Montreal Cognitive Assessment (MoCA) |
| Geriatric Depression Scale (GDS) |
| Instrumental Activities of Daily Living (IADL) |
| Mobile Device Proficiency Questionnaire (MDPQ-16) |
| Computer Proficiency Questionnaire (CPQ) |
| Logical Memory |
| Friendship Scale |
| UCLA Loneliness Scale- Version 3 |
| Quality of Life- AD |
| System Usability Scale |
| Perceived Ease of Use and Usefulness |
| Interpersonal Support Evaluation List |
| Intention Survey |
| Lubben Social Network Index |
| Session Feedback Questions DRAFT |
| Opinion Interview DRAFT |
| Category Fluency |
| Social Activity Frequency (SAQ) |
| Drafts or final copies of all research materials are attached. X Yes |
| 7C. List approximate study dates. Date of IRB approval- August 1, 2024 |
| <b>7D. What is the duration of participants' involvement?</b> Participants' eligibility will be determined |
| following a phone pre-screening and a video screening. If eligible, participants will be randomized into an |



immediate social engagement intervention group or a later intervention group after a 1-hour baseline assessment.

**Group 1 (intervention first)**: Participants in this group will receive 8 weeks of the OneClick social engagement intervention. During this 8-week period, they will be asked to participate in 2 social engagement intervention sessions per week each lasting approximately 45 minutes. A mid-assessment will be done 4 weeks after the beginning of the intervention, and a final post-assessment after 8-weeks of intervention. Both assessments will take 1 hour. Participants will additionally complete a 30-45 minute phone interview at 4 and 8 weeks.

**Group 2 (intervention later):** After being placed in Group 2, participants will receive no planned intervention in the first 8 weeks. They will complete one assessment after 4 weeks and another after 8 weeks. Both sessions will last 1 hour. Then participants will be rolled into the OneClick social engagement intervention lasting 8 weeks. They will complete two additional assessments, one 4 weeks and the other 8 weeks after beginning the video chat intervention These assessments will last 1 hour. Participants will additionally complete a 30-45 minute phone interview at 12 and 16 weeks.

### 7E. How many times will participants engage in research activities?

**Group 1** will complete three assessments: baseline; week 4 post-video chat participation; and week 8 post-video chat participation. They will attend 16 OneClick event sessions.

**Group 2** will complete five assessments: baseline; week 4 after enrollment and before video chat intervention; week 8 after enrollment and before video chat intervention; week 4 post-video chat participation; and week 8 post-video chat participation. They will attend 16 OneClick event sessions.

### 7F. Narratively describe the research procedures in the order in which they will be conducted.

- 1. Phone Pre-Screening: All participants will undergo a phone screening to determine initial eligibility for the next step (video screening). The phone screening will gather information about basic demographics, living arrangements, and visual and auditory acuity. TICS-M will be administered to screen for global cognition. Participants who meet the initial eligibility criteria will be invited to participate in a video screening.
- 2. Informed Consent for Video Screening: Electronic informed consent will be obtained from all participants using REDCap to participate in a screening session over videochat. The participants with MCI will have no deficits in global cognitive functioning, as determined by TICS-M. Subtle cognitive changes observed in these individuals do not impact their ability to provide informed consent; therefore, no proxy consent will be required.
- 3. Video Screening: After obtaining online informed consent, participants will complete a background questionnaire (TSBQ). The Montreal Cognitive Assessment (MoCA) will be administered to assess global cognition. The Geriatric Depression Scale (GDS) will be administered to screen for elevated depressive symptoms. Researchers will review and determine final eligibility for participation. Those who meet eligibility will be invited to participate in the study. If they agree to participate, they will be consented for the intervention study before administering baseline assessment. If a participant does not qualify or prefers not



- to participate despite being eligible, they will be thanked for their participation. The session will last approximately 45 minutes. All participants regardless of eligibility will be paid \$15 for the video screening session.
- 4. Informed Consent for RCT: Electronic informed consent will be obtained from all participants using REDCap for the RCT. Details about the study, expectations, risks, and benefits will be described. All questions will be clarified, and comprehension of the information will be checked by using the teach-back approach. The participants with MCI will have no deficits in global cognitive functioning. Subtle cognitive changes observed in these individuals do not impact their ability to provide informed consent; therefore, no proxy consent will be required.
- 5. Baseline Assessment: Baseline assessment will include participant characterization measures and intervention outcome measures. The session will last approximately one hour.
- 6. Randomization process: The randomization process is designed to achieve appropriate generation of the random allocation sequence and concealment of the allocation sequence. A researcher who is not involved in phone screening, video screening, or informed consent will generate the randomization list prior to the screening of the first person for the randomized, controlled trial. The randomization list will use computer-generated random numbers. The randomization list will be stratified with random permuted blocks. The stratification variable will be Mild Cognitive Impairment (MCI present versus absent). MCI will be defined by a MoCA score of 20-25. The block size will vary randomly between 4 and 6. Research personnel who perform phone screening, video screening, informed consent, or assessments will not be able to access the randomization list. After a potential participant has completed phone screening and video screening, has fulfilled all inclusion criteria, has demonstrated no exclusion criteria, has provided documented informed consent, and has completed baseline assessment, the researcher will unconceal the randomization assignment for the intervention: Group 1 (intervention first) versus Group 2 (intervention later). After assignment, the participant and the researcher who performed informed consent will not be blinded to group allocation.
- 7. Participants in Group 2 will be told they will begin the intervention 8 weeks later and in the meantime will be asked to complete assessments at 4 and 8 weeks after joining the study but before beginning the video chat participation. Participants in Group 1 will be given information about the general research expectations over the next 8 weeks and will be invited to sign up for a technology training session to learn how to use the OneClick system.
- 8. Technology training session: Participants ready to begin the video chat participation will complete a brief technology training session. To help schedule the technology training participants will be contacted by a researcher through their preferred method of communication. Once the technology training is scheduled, participants will be sent a reminder the day prior to their session. A researcher will provide an overview of the purpose and functionality of the OneClick system. A help card will be mailed to the participants with reminders about OneClick login, event sign-up, and participation. It will list a telephone number and email address that can be used for questions or difficulties. One of our research team members will help setup the computer as needed before the 8-week trial if the participant is



- unable to do so with remote instruction. During the training participants will also be provided with an opportunity to RSVP for OneClick video chat events.
- 9. OneClick social engagement intervention: At least two days before starting the intervention, participants will receive a reminder call/email about RSVPing for the OneClick video chat session. If they have not, we will invite them to do so while the researcher is on the phone, in case of difficulties. Participants will receive an email or telephone reminder(s) about the event topic options for the upcoming week and encouraged to sign up for the ones that are of interest to them (no more than 3 reminders will be sent). We will ensure there are at least five unique events that cover a range of topics each week. Each event will last approximately 45 minutes. The event will begin with an introduction to the topic and a set of initial idea for discussion related to the topic. Events include a variety of topics, based on research from a previous study. These topics include arts and culture; nature, health, and wellness; life experiences; science and technology; and recreation and sports. All events include a series of pictures and discussion questions which have been designed to be positive and require a low memory load. Each event will involve a minimum of 3-4 individuals. If an event is not attended by a minimum of 3 participants, we will have a pool of volunteers to join the event who are knowledgeable or interested in the topics to ensure the minimum group size for each event is maintained. Events will be open only to research participants and trained volunteers to ensure a safe and controlled environment for everyone at this stage of product testing and development. During the intervention, we will measure frequency of use, topic selection, discussion duration, and feedback comments/ratings after each event. (i.e. enjoyment, ease of use, quality of video and audio). If participants have not attended an event over the span of a week they will be contacted via their preferred method of communication to remind them to sign up for at least 2 events per week. Participants will be contacted for up to three weeks. If no contact has been made for three weeks, the participant will be dropped from the study and informed via their preferred method of communication.
- 10. Week-4 assessment: 4 weeks after being placed into Group 1 or Group 2, participants will be contacted to schedule a week-4 assessment. Participants in both groups will complete measures related to social connectedness, loneliness, isolation, and quality of life. Group 1 will additionally complete measures related to system usability and perceived enjoyment of the OneClick system. This assessment session will take approximately 1 hour will be administered by a blinded assessor remotely over video or phone. Participants will be informed at the beginning of the assessment not to reveal their group assignment. Both groups will receive \$25 for this session. For Group 1 only, an additional short, semi-structured interview will be administered over video or phone by an unblinded assessor. This will focus on ease of use, usefulness, enjoyment, satisfaction with the topics and conversation, suggestions for updates, and perceptions of social connectedness and will take 30-45 minutes. The interviews will be audiotaped and transcribed verbatim. Group 1 will receive \$15 for completing the interview.



- 11. After this week-4 assessment, a research team member will contact participants in Group 1 to address any questions and issues related to the intervention to help participants remain engaged in the next 4-weeks of intervention.
- 12. Week-8 assessment: 8 weeks after being placed into Group 1 or Group 2, participants will be contacted to schedule a week-8 assessment. Each group's assessment sessions and compensation will be identical to week-4 assessment. This ends Group 1 participation in the study. They will receive a study debriefing and thanked for their time.
- 13. After the week-8 assessment, a research team member will contact participants in Group 2 to schedule their technology training session (described in step #8).
- 14. Group 2 will now begin 8 weeks of video-chat intervention
- 15. Four weeks after completing video chat participation, Group 2 will complete anther assessment. Participants will complete measures related to social connectedness, loneliness, isolation, quality of life, system usability, and perceived enjoyment of the OneClick system. This assessment session will take approximately 1 hour and participants will receive \$25. An additional short, semi-structured interview will be completed over video or phone. This will focus on ease of use, usefulness, enjoyment, satisfaction with the topics and conversation, suggestions for updates, and perceptions of social connectedness and will take 30-45 minutes. The interviews will be audiotaped and transcribed verbatim. Group 2 will receive an additional \$15 for completing the interview. Assessors will no longer be blinded to group assignment.
- 16. Following this assessment, a research team member will contact participants in Group 2 to address any questions and issues related to the intervention to help participants remain engaged in the next 4-weeks of intervention.
- 17. Eight weeks after beginning video chat participation, Group 2 will complete the final assessment. This assessment will follow the exact same procedures and compensation as the assessment done after completing 4 weeks of video chat participation (#15). Group 2 will now end study. They will receive a study debriefing and thanked for their time.

# Section 8. PERFORMANCE SITES TO INCLUDE INTERNATIONAL, SCHOOL, AND COLLABORATIVE STUDIES

| 8A. List <u>all</u> research sites for the protocol. For non-University of Illinois at Urbana-Champaign sites, |
|---|
| describe their status of approval and provide contact information for the site. If the site has an IRB, |
| note whether the IRB has approved the research or plans to defer review to the University of Illinois at |
| Urbana-Champaign. |
| Performances Sites |
| #1 Participant's home |
| #2 UIUC |
| #3 CJE SeniorLife |
| If there are additional performance sites, include them on an attachment and check here: |

| OFFICE FOR THE PROTECTION OF RESEAS | CH SUBJECTS | CTS UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 02/07/2020 |



| 8B. Is this a multi-center study in which the Illinois investigator is the lead investigator, or the |
|---|
| University of Illinois at Urbana-Champaign is the lead site? X Yes No |
| If yes, answer 8C and 8D. If no, proceed to Section 8E. |
| 8C. Who is the prime recipient of funding, if funded? University of Illinois at Urbana-Champaign |
| 8D. What is the management and communication plan for information that might be relevant to the |
| protection of research subjects (e.g. unanticipated problems involving risks to subjects, interim results, |
| and protocol modifications)? This is a multi-site, minimal risk clinical trial and as such will be monitored |
| by an independent Safety Officer. The Principal Investigator (PI) Dr. Wendy Rogers with support from Dr. |
| Raksha Mudar will be responsible for ensuring participants' safety on a daily basis. A Safety Officer (SO) |
| has been appointed to provide data and safety monitoring oversight to monitor participant safety, |
| evaluate the progress of the study, and review procedures for maintaining the confidentiality of data, |
| quality of data collection, management, and analyses. James Graumlich, MD, Associate Chair for |
| Research, Department of Medicine, University of Illinois College of Medicine at Peoria will serve as the |
| SO. Dr. Graumlich has extensive RCT experience. He is an internist with additional training in clinical trial |
| methodology. He has 25 years of experience as a clinical trial investigator, including roles as Principal |
| Investigator of federally-funded research grant protocols. Dr. Graumlich has served as a member of the |
| Data Safety and Monitoring Boards for various clinical trials. |
| No adverse events are expected given that this is a behavioral intervention study of low risk involving use |
| of computer/tablet to engage in conversations with other people over a video chat platform called |
| OneClick. Nevertheless, we do have a protocol in place for documenting and reporting any events to the |
| safety officer (SO). |
| Formal responses to alerts and adverse events will be followed by research staff immediately upon |
| learning about such an event. When an adverse event is identified by a member of the research team, |
| the event will be reported to the PI within 24 hours and recorded on the Adverse Event Form. The |
| University of Illinois will be responsible for maintaining the events forms and submitting reports or summaries to the SO. |
| 8E. If subjects will be recruited from Illinois public or private elementary or secondary schools, |
| additional deadlines and procedures may apply. Criminal background clearances might be required. |
| Special consideration must be given to the exclusion of protected populations. Please contact the |
| School University Research Relations (researchplacements@education.illinois.edu) for more |
| information. Select one: Illinois schools will be used Illinois schools will not be used |
| mileting series and in mileting series with be asea / mileting series with met be asea |

## Section 9. SUBJECT ENROLLMENT GOAL & EQUITABLE SELECTION OF SUBJECTS

| 9A. For each performance site, indicate the estimated total number of participants. | | | | |
|---|---|---|---|---|
| Per | formance Site | # Male | # Female | Total |
| #1 | UIUC | 53 | 53 | 106 |
| #2 | CJE Senior Life | 35 | 35 | 70 |

| OFFICE FOR THE PROTECTION OF RESEAR | CH SUBJECTS | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 02/07/2020 |



| #3 | | | |
|---|---|---|---|
| TOTALS | 88 | 88 | 176 |
| If additional performance sites are included on an a | ttachment, check | here: | |
| 9B. Select all participant populations that will be recruited. | | | |
| Age: | | | |
| Adults (18+ years old) | | | |
| ☐ Minors (≤17 years old) | | | |
| Specific age range, please specify: 65 and older | | | |
| Gender: | | | |
| $\square$ No targeted gender (both men and women will b | | | |
| Targeted gender, please indicate: Men/boys [ | Women/girls | Other, <i>please s</i> | pecify: |
| Race/Ethnicity: | | | |
| $\square$ No targeted race or ethnicity (all races and ethnic | cities will be recrui | ted/included) | |
| Targeted race or ethnicity, please specify: | | | |
| College Students: | | | |
| No targeted college population | | | |
| UIUC general student body | | | |
| Targeted UIUC student population, provide the in | | information, nan | ne of the |
| departmental subject pool, or other specific characte | | | |
| Students at institution(s) other than UIUC, please | | | |
| Any research with students on UIUC's campus needs | to be registered w | ith the <u>Office of t</u> | <u>he Dean of</u> |
| Students. | | | |
| Other: | | | |
| Inpatients | | | |
| Outpatients | | | |
| People who are illiterate or educationally disadva | - | | |
| People who are low-income or economically disa | <u>-</u> | | |
| People with mental or cognitive disabilities or otl | nerwise impaired o | decision-making o | apacities |
| Adults with legal guardians | | | |
| People who are non-English speaking | | | |
| People with physical disabilities | | | |
| Pregnant or lactating women, human fetuses, and/or neonates | | | |
| Prisoners or people with otherwise limited civil freedoms | | | |
| Other, please specify: | | | |
| 9C. Describe additional safeguards included in the p | rotocol to protect | t the rights and w | elfare of the |
| populations selected above. | (2.22) | | |
| We will include older adults with Mild Cognitive Imp | | | |
| Informed Consent. We will mitigate the risks of the f | • | • | |
| highly trained personnel (e.g., graduate student with | · | • | _ |
| older adults or a trained clinician, such as a speech-la | anguage pathologis | st). At UIUC, pers | onnel will be |



supervised by Dr. Mudar who is a clinician by training and has over two decades of experience conducting research involving older adults with cognitive impairment. At CJE, personnel will be supervised by Dr. Danilovich who is also a clinician by training with extensive experience conducting research involving older adults with cognitive impairment. We will make sure to provide encouragement, scheduled breaks, and a supportive environment for the participant. Care will be taken to minimize any feelings of anxiety or discomfort aroused in the participant. Before participants begin assessments, they will be informed that there are no right or wrong answers for the structured interviews or questionnaires. Participants will be informed that if they experience anxiety or discomfort at any point to let us know and we can stop testing immediately. It is important to note that the measures proposed for the study are extensively used for participant testing in the context of studies on aging.

The intervention involves general conversations using the OneClick platform about topics of interest that promote positive reminiscing. We will offer 60 unique events (5/week) that cover a range of topics (e.g., pets; family traditions; baking) that promote reminiscing during conversation, known to produce positive affect in older adults. Participants will be encouraged to sign up for 2 events per week. They will sign up for events of their choosing to minimize feelings of anxiety or discomfort related to any conversation topic. To pre-empt negative experiences of participating in the intervention, especially in participants with MCI, we will provide training to use the OneClick platform, including detailed instructions about participation in the RCT and etiquette for participation, and quick-tip guides to make participation in the intervention enjoyable. We will provide printed materials for reference and contact information in case they require additional help.

### Section 10. INCLUSION/EXCLUSION

# 10A. List specific criteria for inclusion and exclusion of subjects in the study, including treatment and control groups.

Inclusion criteria: Study participants will be adults who are 65 years old and older. All participants will be living independently (i.e., not in assisted living or skilled nursing facilities), fluent in English, and will have adequate visual and auditory acuity to participate. They will have access to a computer or tablet and internet. They will have a Modified Telephone Interview for Cognitive Status (TICS-M) score of 22 or higher, Geriatric Depression Scale (GDS) score of 9 or below.

Additional inclusion criteria for the MCI group include memory complaints objective memory loss measured by a MoCA score of 20-25, and an absence of dementia (no evidence of significant impairment in social or occupational functioning as determined in the background questionnaire).

Exclusion criteria: Potential participants will be excluded if they have a TICS-M score lower than 22 or GDS score higher than 9. They will also be excluded if they have a MoCA score of 19 or less, or if they select "yes" to a diagnosis of Alzheimer's disease or other dementia in the Modified TechSage Background Questionnaire (TSBQ).



| 10B. Explain how the inclusion/exclusion criteria will be assessed and by whom. If special expertise is |
|---|
| required to evaluate screening responses or data, list who will make this evaluation and describe their |
| training and experience. |
| Inclusion/exclusion criteria will be determined by the research team using the screening forms. The |
| research team has sufficient training and experience to carry out the proposed screening. |
| <b>10C. Drafts or final copies of all screening materials are attached.</b> Yes Not Applicable |
| 10D. Describe procedures to assure equitable selection of subjects. Justify the use of the groups |
| marked in Section 9B. Selection criteria that target one sex, race, or ethnic group require a clear |
| scientific rationale. |
| Individuals of both genders will be included with no exclusions made based on racial or ethnic factors. All |
| attempts will be made to recruit equal number of male and female participants. The study will include |
| adults age 65 and older both with and without a diagnosis of MCI. |
| Section 11. RECRUITMENT |
| 11A. Select all recruitment procedures that will be used. |
| Student subject pool, please specify: |
| Email distribution |
| MTurk, Qualtrics Panel, or similar online population, please specify: |
| US Mail |
| ∑ Flyers/brochures |
| Website ad, online announcement (e.g. eWeek), or other online recruitment, please specify: Use of |
| online announcement venues such as eWeek |
| Newspaper ad |
| ∨erbal announcement |
| Other, please specify: Use of Clark-Lindsey Village in-house closed circuit TV system to display |
| electronic flyers. Use of quarterly "President's Letter" including IRB-approved language from recruitment |
| flyer. |
| Not applicable (secondary data only) |
| 11B. Drafts or final copies of all recruitment materials (including verbal scripts) are attached. |
| Yes Not Applicable |
| 11C. For each group of participants, describe the details of the recruitment process. |
| We will use our well-established multi-pronged recruitment strategies, which include word-of-mouth, |
| email, and telephone scripts to members of established registries; flyers and brochures shared by |
| community organizations and partners; advertisements in newspapers and newsletters; and personal |
| visits to community events. All recruitment materials will be pre-approved by the IRB. |
| At UIUC: Participants with and without MCI will be recruited through the I-HELP registry and Dr. Mudar's |
| registry of persons with MCI. The Human Factors and Aging Laboratory directed by Dr. Rogers is part of a |
| consortium that coordinates a registry of potential older research participants through the Beckman |
| Institute at UIUC called I-HELP (Illinois Health and Engagement Lifespan Project). The I-HELP registry |
| module at 5155 canca r rich (minors ricatifi and Engagement Lifespair r toject). The r-rich registry |



currently contains 522 individuals including individuals with a diagnosis of MCI who are interested in participating in university research. Dr. Mudar has a registry of individuals with MCI who are interested in participating in research studies. The MCI registry was developed by Dr. Mudar's research affiliation and ongoing MCI studies with the Carle Neuroscience Institute, which sees approximately 100 MCI patients per year. Additionally, interested participants will be recruited from Carle Neuroscience Institute in collaboration with Dr. Daniel Llano, Staff Neurologist at Carle Hospital.

At CJE: CJE Senior Life supports about 20,000 older adults, which includes individuals with MCI, who live in independent living communities. Participants with and without MCI will be recruited from the 8 retirement community sites managed by CJE SeniorLife as well as their extensions. All sites are independent living. Sites in this study have been purposefully selected throughout the Chicagoland area to reflect a range of racial/ethnic backgrounds to maximize generalizability of findings. Recruitment flyers will be placed in resident mailboxes. Additionally, residents will receive a recruitment flyer during community town-hall meetings.

While general information about the study may be given in community settings, all formal recruitment will be completed via telephone to ensure privacy and individual service. The research team will complete encounter forms for all potential participants. The team will document all attempts to contact participants and will vary day and time of contact attempts if the participant is not reachable on the first attempt. During the recruitment pre-screening call, the research staff will follow a script to gather information about eligibility status and give information about the study. The research staff will clearly explain the time commitment, expectations for participation, and answer any questions the participant asks. If the person is eligible and expresses interest in enrolling, the team will schedule an appointment for obtaining informed consent and enrolling the participant in the study. If the person is ineligible, staff will follow a script to provide this information.

### Section 12. REMUNERATION AND PLAN FOR DISTRIBUTION

| Refer to the University <u>Business and Financial Policies and Procedures</u> for further guidance on the |
|---|
| compensation process and reporting requirements. |
| 12A. Will subjects receive inducements or rewards before, during, or after participation? |
| ∑ Yes ☐ No |
| If yes, complete the rest of Section 12. If no, proceed to Section 13. |
| 12B. Select all forms of remuneration that apply. |
| Cash, please specify amount: |
| Check, please specify amount: |
| Gift Certificate, please specify amount: All participants who complete a video screening session will |
| receive \$15 Amazon e-code. To promote the highest retention rate possible in the RCT, participants will |
| be compensated \$25 at each assessment session. There is an additional supplemental interview that will |
| be given to participants currently receiving the intervention and they and will be paid \$15 for each |
| supplemental interview. Although participants in Group 2 will complete two additional assessments |



| (week-12 and week-16), they will be compensated for these two additional assessments. Also, participants will be allowed to keep their OneClick subscription for a year free of cost. |
|---|
| □ Lottery, please specify amount: and odds: □ Course Credit, please specify amount: and specify equivalent alternative activity: □ Other, please specify: Amazon e-codes will be the primary form of payment, but participants can request an alternative method (cash or check). |
| 12C. Will payment be prorated before, during, or after participation? ☐ Yes, please specify how: In the event participants withdraw from the study early, they will receive payment for any assessments they have completed. ☐ No |
| 12D. For each group of participants, describe the details of the remuneration plan, including how, |
| when Payments (Amazon gift card; checks; cash) will be distributed at the end of the study, or at the end of participation, determined by a researcher. Participants will receive a check by mail or an Amazon E-code via email depending upon their preference. |
| 12E. The information listed above is provided on the relevant consent forms. Yes |

### Section 13. RISKS & BENEFITS

13A. Describe all known risks to the participants for the activities proposed, such as risks to the participants' physical well-being, privacy, dignity, self-respect, psyche, emotions, reputation, employability, and criminal and legal status. Risks must be described on consent forms.

There are no specific physical or psychological risks associated with cognitive, psychological, or usability assessments in this research. The assessments include outcome measures that have been used previously with this population, including technology evaluations in persons with MCI, by the investigators. The primary risks of the evaluations and observations are fatigue and frustration due to the difficulty of some tasks. The potential risks for using a novel social engagement platform (small group video discussion) is hesitation in interacting with strangers.

### 13B. Describe the steps that will be taken to minimize the risks listed above.

To reduce the risks of fatigue and frustration, we will provide encouragement, scheduled breaks, and a supportive environment to make participation an interesting and beneficial experience. The events will be initiated by a host, a member of our research team. Afew conversational prompts will be provided to facilitate interactions. Also, participants will have the options to only sign up for topics of their choice. Our prior research has shown that older adults form new friendships (i.e., with strangers) when they coparticipate in an activity and/or share interests. OneClick, the social platform under investigation, is designed to connect people over shared interests.



| 13C. Indicate the risk level. |
|---|
| No more than minimal risk |
| (The probability and magnitude of harm or discomfort anticipated for participation in the proposed |
| research are not greater in and of themselves than those ordinarily encountered in daily life or during |
| the performance of routine physical or psychological examinations or tests). |
| More than minimal risk (answer 13D) |
| 13D. If you checked that the research is more than minimal risk, describe the provisions for monitoring |
| the data to ensure the safety of subjects, such as who will monitor data and how often, what criteria |
| will be used to stop the research, etc. |
| • |
| 13E. Describe the expected benefits of the research to the subjects and/or to society. |
| The findings from this study will have major implications on the launch and commercialization of a novel |
| Internet-based social engagement platform for older adults with and without MCI. Furthermore, by |
| making the platform accessible for these specific user groups, OneClick also will become more accessible |
| to other, non-impaired and younger, users. This is the promise and benefit of universal, user-centered |
| design. The platform could offer an easy, affordable (i.e., free) socialization avenue especially to people |
| living in remote, socially-isolated areas and to those feeling socially isolated and lonely. The direct |
| benefits to the participants and society outweigh any potential risks incurred through participation. |
| benefits to the participants and society outweight any potential risks incurred through participation. |
| 13F. Weigh the risks with regard to the benefits. Provide evidence that benefits outweigh risks. |
| We have taken precautions to decrease foreseeable potential risks to the participants as a result of their |
| participation in this study. Overall the risks of interacting with the OneClick system, participating in the |
| interview and completing the questionnaires should be minimal. A potential benefit for the participants |
| is social and cognitive stimulation. These benefits outweigh the potential risks, which are minimal to |
| begin with and will be further minimized by the proposed research. |
| begin with and win be farther minimized by the proposed research. |
| Costing 14 INFORMED CONSENT PROCESS TO INCLUDE, WAIVERS ASSENTS ALTERATIONS FTC |
| Section 14. INFORMED CONSENT PROCESS TO INCLUDE: WAIVERS, ASSENTS, ALTERATIONS, ETC. |
| 14A. Indicate all that apply for the consent/assent/parental permission process. |
| Written informed consent (assent) with a document signed by |
| □ adult subjects □ parent(s) or guardian(s) □ adolescents aged 8–17 years |
| Waiver of Documentation (signature) of Informed Consent (include the relevant Waiver Form) |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| Waiver of Informed Consent (include the relevant Waiver Form) |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| Alteration of Informed Consent (include the relevant Alteration Form) |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| 14B. List all researchers who will obtain consent/assent/parental permission from participants. |



| Wendy A. Rogers, Raksha Mudar, George Mois, Elizabeth Lydon, Vincent Mathias (For more information |
|---|
| of the researchers, please see attached research team form). |
| 14C. Describe the method for obtaining consent/assent/parental permission. Informed consent will be |
| obtained online before any testing is undertaken. Details related to the study will be discussed at length. |
| Any questions pertaining to the study and participation will be answered. The online informed consent |
| process will be administered over REDCap with a research team member and signed electronically. |
| Participants will receive a copy of the signed document for their records (either electronically or a paper |
| version mailed to their home). |
| 14D. Describe when consent/assent/parental permission will be obtained. Informed consent for the |
| video screening will be obtained before the video screening session begins. Informed consent for the RCT |
| will be obtained before the baseline assessment session begins. |
| 14E. Will participants receive a copy of the consent form for their records? |
| Yes No, if no, explain: |
| 14F. Indicate factors that may interfere or influence the collection of voluntary informed |
| consent/assent/parental permission. |
| No known factors |
| Research will involve students enrolled in a course or program taught by a member of the research |
| team |
| Research will involve employees whose supervisor(s) is/are recruiting participants |
| Participants have a close relationship to the research team |
| Other, specify any relationship that exists between the research team and participants: |
| If applicable, describe the procedures to mitigate the above factors. |
| <b>14G. Copies of the consent form(s) are attached.</b> $\boxtimes$ Yes $\square$ Not applicable |
| 14H. Will this project be registered as a clinical trial? X Yes No |
| If yes, effective January 21, 2019, an informed consent form must be posted on the Federal Web site |
| after the clinical trial is closed to recruitment, and no later than 60 days after the last study visit. |
| Section 15. DEVICES & DRUGS |
| Indicate if your research includes any of the following. |
| Equipment [Researchers collecting physiological data, not testing the device] |
| (include Appendix A, the <u>Research Equipment Form</u> ) |
| Devices [Researchers planning to test devices on human subjects] |
| (include Appendix B, the <u>Device Form</u> ) |
| Materials of Human Origin |
| (include Appendix C, the <u>Biological Materials Form</u> ) |
| ☐ Drugs and Biologics |
| (include Appendix D, the <u>Drug and Chemical Usage Form</u> ) |



| | MRI AT BIC To use the <u>Beckman Institute Biomedical Imaging Center</u> (BIC) in human subject's |
|---|---|
| | research, you must obtain prior approval from the BIC (217.244.0446; <a href="mailto:ryambert@illinois.edu">ryambert@illinois.edu</a> ) and use |
| | BIC-approved screening and consent forms. Attach: |
| | ☐ BIC approval ☐ BIC screening form ☐ BIC consent form |
| | Section 16. CONFIDENTIALITY OF DATA & PRIVACY OF PARTICIPATION |
| | 16A. How is participant data, records, or specimens identified when received or collected by |
| | researchers? Identifiers include, but are not limited to, name, date of birth, email address, street |
| | address, phone number, audio or video recordings, and SSN. |
| | No identifiers are collected |
| | Direct identifiers are collected |
| | $\square$ Indirect identifiers (e.g. a code or pseudonym used to track participants); |
| | Does the research team have access to the identity key? $igtigtigthedown$ Yes $igsqcup$ No |
| | 16B. Select all methods used to safeguard research records during storage: |
| | $oxed{oxed}$ Written consent, assent, or parental permission forms are stored separately from the data |
| | Data is collected or given to research team without identifiers |
| | Data is recorded by research team without identifiers |
| | Direct identifiers are removed from collected data as soon as possible |
| | Direct identifiers are deleted and no identity key exists as soon as possible |
| | Participant codes or pseudonyms are used on all data and the existing identity key is stored |
| | separately from the data |
| | Electronic data is stored in a secure, <u>UIUC-approved location</u> , <i>please specify</i> PHI Box |
| | Hard-copy data is stored in a secure location on UIUC's campus, please specify |
| | Other, please specify: |
| | <b>16C. How long will identifiable data be kept?</b> Electronic versions of the data will be archived on PHI box |
| | <b>16D. Describe provisions to protect the privacy interests of subjects.</b> Information about this research |
| | study will remain confidential unless we are required by law to release it. Electronic copies of the signed |
| | consent forms will be stored on PHI box. All participants will be assigned a participant code that is not |
| | related to their personal information in any way. This participant code will be used for all data collection. |
| | There will be one master sheet linking participant name to participant code. This sheet will be |
| | electronically stored on the PHI box with restricted access to the research team. Allelectronic copies of |
| | the data will be stored by study ID in the PHI box that only the research team has access to including the |
| | audio recordings. Once audio files are uploaded to the PHI box, these files will be deleted from the initial |
| | recording device. Strict security will be maintained to access the PHI box. No identifying information will |
| | be mentioned in any presentations or publications. Similar procedures at these study sites have proven |
| | to effectively prevent loss of confidentiality. |
| | 16E. Describe the training and experience of all persons who will collect or have access to the data. |
| | Data collection will be carried out by trained personnel and access to study data will be limited to |
| ı | researchers directly involved with this research study who have been trained in methods to protect the |



confidentiality, including IRB CITI training requirements. Workshops are held to ensure that all individuals involved in research keep their certification current.

| Section 17. | DISSEMINATION | OF | RESU | LTS |
|-------------|---------------|----|------|-----|
|-------------|---------------|----|------|-----|

| 17A. List proposed forms of dissemination (e.g. journal articles, thesis, academic paper, conference |
|---|
| presentation, sharing within industry, etc.). |
| Results may be disseminated in the following forms: journal articles, thesis or academic papers, |
| conference proceedings and presentations, and technical reports. |
| 17B. Will any identifiers be published, shared, or otherwise disseminated? 🗌 Yes 🔀 No |
| If yes, does the consent form explicitly ask consent for such dissemination, or otherwise inform |
| participants that it is required in order to participate in the study? Yes |
| 17C. Do you intend to put de-identified data in a data repository? 🔀 Yes 🗌 No |
| If yes, explain how data will be de-identified. |
| We will use subject ID to substitute the real name of the participants. |
| Section 18. INVESTIGATOR & DEPARTMENTAL ASSURANCES |
| <ul> <li>I certify that the information provided in this application is complete and correct.</li> </ul> |
| <ul> <li>I certify that I will follow my IRB Approved Protocol.</li> </ul> |
| <ul> <li>I accept ultimate responsibility for the conduct of this study, the ethical performance of the</li> </ul> |
| project, and the protection of the rights and welfare of the human subjects who are directly or |
| indirectly involved in this project. |
| <ul> <li>I will comply with all applicable federal, state and local laws regarding the protection of human</li> </ul> |
| subjects in research. |
| <ul> <li>I will ensure that the personnel performing this study are qualified and adhere to the provisions</li> </ul> |
| of this IRB-certified protocol. |
| The original signature of the PI is required before this application may be processed (electronic |
| signatures are acceptable). |
| (SIAPON) |
| 8/2/22 |
| Principal Investigator Date |
| If the PI is not eligible to serve as PI under the Campus Administrative Manual, the applicable |
| academic dean, institute director, or campus administrative officer indicates their approval of the |
| researcher to act as Principal Investigator. Please note that departmental assurance only needs to be |
| provided in the initial application. |



| Name of Authorizing Individual | |
|-------------------------------------|----------|
| Signature of Authorizing Individual | <br>Date |



### **Video Technology-based Social Engagement**

You are being asked to participate in a voluntary research study. The purpose of this study is to evaluate a video chat technology called OneClick. In distinct contrast to existing social media and online chat, dating, or meet-up applications, OneClick connects people virtually for an indepth, meaningful conversation on topics they are passionate about. No exchange of private information or physical meeting is required.

## **University of Illinois Urbana-Champaign**

**Principal Investigator Name:** Wendy A. Rogers, Ph.D.

Department and Institution: Kinesiology and Community Health, College of Applied Health

Sciences, University of Illinois Urbana-Champaign Contact Information: Phone – (217) 300-5445 Sponsor: The National Institute on Aging

## Why am I being asked?

You are being invited to take part in this research study because you are 65 years or older and have completed the phone and video screening processes. Approximately 120 subjects may be involved in this research.

Your participation in this research is voluntary. If you decide to participate, you are free to withdraw at any time.

### What procedures are involved?

This study first involves completing preliminary assessments over video chat including information about demographics, your preferences on technology, your memory, and other questionnaires about your social networks, mental health, and wellbeing. This assessment is expected to take one hour. After completing these assessments, you will be randomized to participate in the intervention immediately (Group 1) or later (Group 2).

**If you are put in Group 1**, you will be asked to schedule a technology training session to learn to use the OneClick system.

<u>Technology Training</u>: Training involves viewing an instructional video that provides an overview of the OneClick system and steps to use it. You will then have the opportunity to ask questions and to explore the OneClick system. This process will take 30-60 minutes. To help schedule the technology training you will be contacted by a researcher through your preferred method of communication. Once the technology training is scheduled we will provide you reminders prior to the scheduled date.



<u>Video chat Participation</u>: After technology training, you will be invited to sign up for events on OneClick. You are expected to attend 2 video chat events of your choice per week for 8 weeks. Each video chat event will last 30-45 minutes. You can select which events you prefer to attend based on your interests and sign up via an online calendar. In the event, you will see a short slide presentation about the topic of interest. After the slide show, you go into a virtual breakout room to have a casual conversation with others about the topic. Ideas for conversation will be shared. You will be asked to keep confidential any information shared during these conversations.

We will provide you with reminders about the events you have signed up for and links to the RSVP page which will allow you to select events on an ongoing basis. These reminders will provide you with contact information to receive any assistance that you might need with the RSVP process. If you do not attend any sessions for more than three weeks in a row, you may be withdrawn from the study.

<u>Week 4 Post-Video Chat Participation Assessment:</u> At approximately 4 weeks from the start of your participation in events, researchers will contact you to participate in a Week 4 assessment conducted over OneClick. During this assessment you will complete some questionnaires. Assessment is expected to take 1 hour. In addition, you will be asked to complete a short interview over video or phone to provide your initial feedback on using the OneClick system. The interview is expected to take 30-45 minutes.

<u>Week 8 Post-Video Chat Participation Assessment</u>: Once you have completed your 8 weeks of participation, researchers will contact you to complete a Week 8 assessment conducted over OneClick. The assessment is approximately 1 hour long. During this assessment you will complete some questionnaires, and you will again be asked to participate in a 30-45 minute interview over video or phone to provide feedback on your experience. At this point, your participation is complete and you will be paid, debriefed, and thanked for your participation in the study.

If you are put into Group 2, you will complete two assessments at approximately 4 and 8 weeks from today's date. Researchers will schedule these assessments to complete over OneClick. Each assessment is expected to take 1 hour. During these assessments you will complete some questionnaires. After 8 weeks, you will be asked to schedule a technology training session to learn how to use the OneClick system and will be invited to participate in 8 weeks of OneClick events.

<u>Technology Training</u>: Training involves viewing an instructional video that provides an overview of the OneClick system and steps to use it. You will then have the opportunity to ask questions and to explore the OneClick system. This process will take 30-60 minutes. To help schedule the technology training you will be contacted by a researcher through your preferred method of



communication. Once the technology training is scheduled we will provide you reminders prior to the scheduled date.

<u>Video Chat Participation</u>: After technology training, you will be invited to sign up for events on OneClick. You are expected to attend 2 video chat events of your choice per week for 8 weeks. Each video chat event will last 30-45 minutes. You can select which events you prefer to attend based on your interests and sign up via an online calendar. In the event, you will see a short slide presentation about the topic of interest. After the slide show, you go into a virtual breakout room to have a casual conversation with others about the topic. Ideas for conversation will be shared. You will be asked to keep confidential any information shared during these conversations.

We will provide you with reminders about the events you have signed up for and links to the RSVP page which will allow you to select events on an ongoing basis. Furthermore, these reminders will provide you with contact information to receive any assistance that you might need with the RSVPing process. If you do not attend any sessions for more than three weeks in a row, you may be withdrawn from the study. If you do not attend any sessions for more than three weeks in a row, you may be withdrawn from the study.

<u>Week 4 Post-Video Chat Participation Assessment</u>: Once you have completed 4 weeks of participation in events, researchers will contact you to participate in this assessment conducted over OneClick. During this assessment you will complete some questionnaires. Assessment is expected to take 1 hour. In addition, you will be asked to complete a short interview over video or phone to provide your initial feedback on using the OneClick system. The interview is expected to take 30-45 minutes.

<u>Week 8 Post-Video Chat Participation Assessment:</u> Once you have completed your 8 weeks of participation in OneClick events, researchers will contact you to complete this assessment. The assessment is approximately 1 hour long. During this assessment you will complete some questionnaires, and you will again be asked to participate in a 30-45 minute interview over video or phone to provide feedback on your experience. At this point, your participation is complete and you will be paid, debriefed, and thanked for your participation in the study.

### What are the potential risks and discomforts?

There are no specific physical or psychological risks associated with the assessments in this research. The primary risks of the assessments and observations are fatigue and frustration due to the difficulty of some tasks. We will provide encouragement, scheduled breaks, and a supportive environment to make participation an interesting and beneficial experience. There are no known risks of participating in a discussion other than the initial uneasiness of talking to strangers. However, given that the topics chosen are of mutual interests and the host will open the discussion, the uneasiness will be minimized.





## Are there benefits to participating in the research?

You are not likely to benefit directly from this study other than having an opportunity to socially engage in topic-centered conversations with others. The findings from this study will have implications for making video chat technology more accessible to older adults both with and without memory complaints.

## What other options are there?

By law, participation in research is completely **voluntary** and may be stopped at any time without question or negative consequence. Because this is not a treatment study, there are no alternatives to participation other than the termination of involvement in the study.

## Will my study-related information be kept confidential?

We will use all reasonable efforts to keep your personal information confidential, but we cannot guarantee absolute confidentiality. When this research is discussed or published, no one will know that you were in the study. But, when required by law or university policy, identifying information may be seen or copied by: a) The Institutional Review Board that approves research studies; b) The Office for Protection of Research Subjects and other university departments that oversee human subjects research; c) University and state auditors responsible for oversight of research; d) Federal regulatory agencies such as the Office of Human Research Protections in the Department of Health and Human Services; or e) The National Institute on Aging.

The data collected in this study will be de-identified and put into an archived repository and stored on a secure server. The link between your name and code will be kept in a password-protected file and will be maintained by the registry coordinator. This link will be used to match and share your data if you are determined to be eligible to participate.

We will ask everyone in the group discussion to respect the privacy of other participants and to treat anything said in the group as confidential. However, please remember there is no guarantee that other participants will abide by that request.

### Will I be reimbursed for any expenses or paid for my participation in this research?

You will receive \$25 for completing the assessment sessions over OneClick. You will also receive \$15 for completing the interviews over the phone. You will receive your payment via Amazon ecode or another method upon request. You will also have continued access to OneClick for one year free of cost. If you do not finish an assessment session, you will receive compensation for the number of sessions completed.

### Can I withdraw or be removed from the study?

If you decide to participate, you are free to withdraw your consent and discontinue participation at any time. If you decide to withdraw your consent and discontinue participation,

ILLINOIS IRB APPROVED

the researchers will ask you to complete a very short termination visit over the phone or video chat. The researchers also have the right to stop your participation in this study without your consent if they believe it is in your best interests.

### Will data collected from me be used for any other research?

Some of the tests that are performed in this research study are used in other studies by the University of Illinois Urbana-Champaign. We have established a data repository that can store the results of your participation in these tests with your permission to be studied in future projects. Please note that the data that are stored are given a unique identification code so that none of the data are able to be identified. Only the researcher and approved personnel will have access to the identification code key.

## Who should I contact if I have questions?

If you have questions about this project, you may contact Wendy Rogers at <a href="wendyr@illinois.edu">wendyr@illinois.edu</a>. If you have any questions about your rights as a participant in this study or any concerns or complaints, please contact the University of Illinois Urbana-Champaign Office for the Protection of Research Subjects at 217-333-2670 or via email at <a href="irb@illinois.edu">irb@illinois.edu</a>. A copy of this consent form will be mailed or emailed to you for your records.

I certify that I am 18 years old or older. I certify that I have read and understand the information in the above consent. I indicate my willingness to voluntarily participate in this study by typing my name in the box below. I understand that this is equivalent to signing a physical document.

| Particip | ant Name (type | your name here): |
|----------|----------------|------------------|
| Date: | | |

**SUBMIT** 



IRB Number: 22212

IRB Approval Date: 08/11/2022 IRB Expiration Date: 9/14/2026



### **Video Technology-based Social Engagement**

You are being asked to complete a video screening to determine your eligibility for a voluntary research study. The purpose of this study is to investigate the benefits of using a new video chat technology called OneClick. This is a less than minimal risk study and there is no direct benefit to you for participating.

**University of Illinois Urbana-Champaign** 

**Principal Investigator Name:** Wendy A. Rogers, Ph.D.

Department and Institution: Kinesiology and Community Health, College of Applied Health

Sciences, University of Illinois Urbana-Champaign Contact Information: Phone – (217) 300-5445

**Sponsor**: The National Institute on Aging

### Why am I being asked?

You are being invited to take part in this research study because you are 65 years or older and have completed the phone screening process.

Your participation in this research is voluntary. If you decide to participate, you are free to withdraw at any time.

### What procedures are involved?

This video screening involves a brief memory test and some questionnaires. This video screening is expected to take 30-45 minutes. Once completed, this will determine your eligibility to participate in an intervention study on video technology-based social engagement.

If you meet the eligibility for the study, you will be invited to participate in a study on video technology-based social engagement using OneClick. You will go through an additional informed consent process detailing the full study procedures. If you do not wish to participate, you are able to decline participation at any point. You will be paid for your time in the study.

In some cases, eligibility for the study will need to be reviewed by the Principal Investigators and research team. If this is the case, at the end of the video screening we will let you know that we need time to determine eligibility. We will follow-up with you over phone or email once your eligibility is determined.

If you are not eligible for the study, you will be paid and asked if you would like to be added to our database for future study participation.

### What are the potential risks and discomforts?

There are no specific physical or psychological risks associated with the assessments in this

ILLINOIS
IRB APPROVED

IRB Number: 22212 IRB Approval Date: 09/15/2021

IRB Expiration Date: 9/14/2026



research. The primary risks of the assessments and observations are fatigue and frustration due to the difficulty of some tasks. We will provide encouragement, breaks, and a supportive environment to make participation an interesting and beneficial experience. There are no known risks of participating in the video screening.

### Are there benefits to participating in the research?

You are not likely to benefit directly from this video screening study. The findings from this screening will determine if you are eligible to participate in the intervention study.

### What other options are there?

By law, participation in research is completely **voluntary** and may be stopped at any time without question or negative consequence. Because this is not a treatment study, there are no alternatives to participation other than the termination of involvement in the study.

### Will my study-related information be kept confidential?

We will use all reasonable efforts to keep your personal information confidential, but we cannot guarantee absolute confidentiality. When this research is discussed or published, no one will know that you were in the study. But, when required by law or university policy, identifying information may be seen or copied by: a) The Institutional Review Board that approves research studies; b) The Office for Protection of Research Subjects and other university departments that oversee human subjects research; c) University and state auditors responsible for oversight of research; d) Federal regulatory agencies such as the Office of Human Research Protections in the Department of Health and Human Services; or e) The National Institute on Aging.

The data collected in this study will be de-identified and put into an archived repository and stored on a secure server. The link between your name and code will be kept in a password-protected file and will be maintained by the registry coordinator. This link will be used to match and share your data if you are determined to be eligible to participate.

### Will I be reimbursed for any expenses or paid for my participation in this research?

You will be compensated \$15 for your participation in the video screening via Amazon E-Code or an alternative method upon request.

## Can I withdraw or be removed from the study?

If you decide to participate, you are free to withdraw your consent and discontinue participation at any time. The researchers also have the right to stop your participation in this study without your consent if they believe it is in your best interests.

ILLINOIS
IRB APPROVED



### Will data collected from me be used for any other research?

Some of the tests that are performed in this research study are used in other studies by the University of Illinois Urbana-Champaign. We have established a data repository that can store the results of your participation in these tests with your permission to be studied in future projects. Please note that the data that are stored are given a unique identification code so that none of the data are able to be identifiable. Only researchers and approved personnel will have access to the identification code key.

## Who should I contact if I have questions?

If you have questions about this project, you may contact Wendy Rogers at <a href="wendyr@illinois.edu">wendyr@illinois.edu</a>. If you have any questions about your rights as a participant in this study or any concerns or complaints, please contact the University of Illinois Urbana-Champaign Office for the Protection of Research Subjects at 217-333-2670 or via email at <a href="irb@illinois.edu">irb@illinois.edu</a>.

A copy of this consent form will be mailed or emailed to you for your records.

I certify that I am 18 years old or older. I certify that I have read and understand the information in the above consent. I indicate my willingness to voluntarily participate in this study by typing my name in the box below. I understand that this is equivalent to signing a physical document.

| Particip | ant Name (type | your name here): |
|----------|----------------|------------------|
| Date: | | |

**SUBMIT** 





## **Research Team**

For Listing Additional Researchers who are Involved in the Project All forms must be typewritten and submitted via email to irb@illinois.edu.

When to use this form: If there are collaborating researchers participating in a research study, including those from other institutions, complete this form by listing all collaborating researchers. Include all persons who will be: 1) directly responsible for project oversight and implementation, 2) recruitment, 3) obtaining informed consent, or 4) involved in data collection, analysis of identifiable data, and/or follow-up. Please copy and paste text fields to add additional research team members.

Note:

- Changes made to the Principal Investigator require a revised <u>Protocol Form</u> and an <u>Amendment</u> Form.
- A complete Research Team form with all research team members included needs to be submitted every time the research team is updated.

### **Section 1. PROTOCOL INFORMATION**

| 1A. Principal Investigator: Dr. Wendy Rogers |
|-------------------------------------------------------------|
| 1B. Protocol Number: 22212 |
| 1C. Project Title: Video Technology-based Social Engagement |

### **Section 2. ADDITIONAL INVESTIGATORS**

| Full Name: Raksha Mudar | Degree: PhD | | Dept. or Unit: Applied |
|---|---|---|---|
| | | | Health Sciences - SHS |
| Professional Email: raksha@illinois.edu | | Phone: 2 | 17-333-4718 |
| Campus Affiliation: | | | |
| igwedge University of Illinois at Urbana-Champaign $igwdot$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔲 Un | dergradua | te Student |
| Visiting Scholar Other, please specify: | _ | | |
| Training: | | | |
| Required CITI Training, Date of Completion (valid with | in last 3 years) | : 07/29/20 | 22 |
| Additional training, <b>Date of Completion</b> : | | | |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study prod | edures 🔀 Har | ndling ider | ntifiable data |
| Other, please specify: project oversight | | | |
| If administering biomedical study procedure (e.g., blood draws, scans, depression index, etc.), please | | | |
| specify the procedure(s): | | | |
| This researcher should be copied on OPRS and IRB correspondence. | | | |
| This researcher is no longer an active research team member. | | | |



# of Research Subjects Research Team

| te added to research team: 07/26/2021 Date removed from research team: | | |
|---|---|---|
| Full Name: Elizabeth Lydon | Degree: M.S. | Dept. or Unit: Applied |
| | | Health Sciences- SHS |
| Professional Email: elydon2@illinois.edu | | Phone: 217-265-6574 |
| Campus Affiliation: | | |
| ☐ University of Illinois at Urbana-Champaign ☐ Other, p | olease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate Student Undergraduate Student | | |
| Visiting Scholar Other, please specify: | | |
| Training: | | |
| Required CITI Training, Date of Completion (valid with | in last 3 years): | 06/29/2021 |
| Additional training, <b>Date of Completion:</b> | | |
| Role on Research Team (check all that apply): | | |
| ig Recruiting $ig $ Consenting $ig $ Administering study produced | cedures 🔀 Han | dling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, e | tc.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | rrespondence. | |
| This researcher is no longer an active research team r | member. | |
| Date added to research team: 07/26/2021 | Date removed | from research team: |
| Full Name: Shraddha Shende | Degree: M.S. | Dept. or Unit: Applied |
| | | Health Sciences- SHS |
| Professional Email: sshende2@illinois.edu | | Phone: 217-265-6574 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Other, p | olease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate S | Student 🗌 Und | ergraduate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid within last 3 years): 8/27/2022 | | |
| Additional training, <b>Date of Completion</b> : | | |
| Role on Research Team (check all that apply): | | |
| Recruiting Consenting Administering study prod | cedures 🔀 Han | dling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB correspondence. | | |
| OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS | UNIVERSITY OF ILLINOIS | S AT URBANA-CHAMPAIGN |

805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333-2670 irb@illinois.edu www.irb.illinois.edu Revised: 4/19/2021

2 of 18



## **Research Team**

| This researcher is no longer an active research team member. | | | |
|---|---|---|---|
| Date added to research team: 07/26/2021 | Date removed from research team: | | |
| Full Name: Madina Khamzina | Degree: MPH | | Dept. or Unit: Applied<br>Health Sciences-<br>Community Health |
| Professional Email: madinak2@illinois.edu | Phone: 217-300-5445 | | |
| Campus Affiliation: | | | |
| University of Illinois at Urbana-Champaign Other, p | lease specify: | | |
| Campus Status: | | | |
| ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S | Student 🔲 Un | dergradua | ate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | | |
| Training: | | | |
| ig Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | : 06/30/20 | 020 |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| $ig igselow{igselow}{igselow}$ Recruiting $igotimes$ Consenting $igotimes$ Administering study proc | edures 🔀 Hai | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, ( | etc.), plea | se specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | • | | |
| This researcher is no longer an active research team n | | | |
| Date added to research team: 07/26/2021 Da | ite removed fr | om resea | rch team: 12/15/2021 |
| | | | T. |
| Full Name: Allura Lothary | <b>Degree:</b> PhD | | Dept. or Unit: Applied |
| | | | Health Sciences- |
| | | | Community Health |
| Professional Email: alothary@illinois.edu | <b>Phone:</b> 217-300-5445 | | |
| Campus Affiliation: | | | |
| $\bigsqcup_{-}$ University of Illinois at Urbana-Champaign $\bigsqcup_{-}$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate Student Undergraduate Student | | | |
| Visiting Scholar Other, please specify: Postdoctoral | Research Asso | ciate | |
| Training: | | 40/05/2 | 222 |
| Required CITI Training, <b>Date of Completion</b> (valid within | in last 3 years) | : 10/05/20 | 020 |
| Additional training, <b>Date of Completion</b> : | | | |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study procedures Handling identifiable data | | | |
| Other, please specify: | | | |

OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN

805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333-2670 irb@illinois.edu www.irb.illinois.edu Revised: 4/19/2021



## **Research Team**

| If administering biomedical study procedure (e.g., blood procedure(s): | draws, scans, o | etc.), plea | se specify the |
|---|---|---|---|
| This researcher should be copied on OPRS and IRB co | respondence. | | |
| This researcher is no longer an active research team n | nember. | | |
| Date added to research team: 07/26/2021 Da | ite removed fr | om resea | rch team: 09/10/2021 |
| Full Name: Saahithya Gowrishankar | Degree: B.S. | | Dept. or Unit: Applied Health Sciences- Community Health |
| Professional Email: sg14@illinois.edu | Phone: 2 | | 17-300-5445 |
| Campus Affiliation: | | | |
| <ul> <li>☑ University of Illinois at Urbana-Champaign ☐ Other, please specify:</li> <li>Campus Status:</li> <li>☐ Faculty ☑ Academic Professional/Staff ☐ Graduate Student ☐ Undergraduate Student</li> <li>☐ Visiting Scholar ☐ Other, please specify:</li> </ul> | | | |
| Training: ☐ Required CITI Training, Date of Completion (valid within) ☐ Additional training, Date of Completion: | in last 3 years) | : 05/29/20 | 019 |
| Role on Research Team (check all that apply): | | | |
| ig Recruiting $ig $ Consenting $ig $ Administering study proc | edures 🔀 Hai | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | respondence. | | |
| This researcher is no longer an active research team n | nember. | | |
| Date added to research team: 07/26/2021 Date | ate removed f | rom resea | arch team: 04/08/2022 |
| Full Name: Sarah Jones | Degree: | | <b>Dept. or Unit:</b> Applied Health Sciences- SHS |
| Professional Email: sarahej3@illinois.edu | Phone: 2 | | 217-265-6574 |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: | | dergradua | ate Student |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid within last 3 years): 08/01/2022 | | | |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| $oxed{\boxtimes}$ Recruiting $oxed{\boxtimes}$ Consenting $oxed{\boxtimes}$ Administering study procedures $oxed{\boxtimes}$ Handling identifiable data | | | |



## **Research Team**

| Other, please specify: | | |
|---|---|---|
| If administering biomedical study procedure (e.g., blood | draws scans etc.) nle | ase specify the |
| procedure(s): | diaws, scalis, etc.,, pic | ase specify the |
| This researcher should be copied on OPRS and IRB co | prrospondonco | |
| This researcher is no longer an active research team | | |
| Date added to research team: 07/26/2021 Date removed from research team: | | |
| - un | T | T |
| Full Name: Ari Sovsic | Degree: | Dept. or Unit: Applied |
| | 1 | Health Sciences- SHS |
| Professional Email: asovsi2@illinois.edu | Phone: | 217-265-6574 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Uther, | please specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate | Student 🔀 Undergradu | ate Student |
| Visiting Scholar Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | nin last 3 years): 08/28/2 | 2019 |
| Additional training, Date of Completion: | | |
| Role on Research Team (check all that apply): | | |
| ig Recruiting $ig $ Consenting $ig $ Administering study pro | cedures 🔀 Handling ide | entifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, etc.), ple | ase specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | orrespondence. | |
| This researcher is no longer an active research team | member. | |
| Date added to research team: 08/31/2021 | Date removed from rese | arch team: 05/03/2022 |
| Full Name: Kelly Kepka | Degree: | Dept. or Unit: Applied |
| Tan name weny wepwa | 3-58. 5-5. | Health Sciences- MCB |
| Professional Email: kepka2@illinois.edu | Phone: | 217-300-5445 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Other, | nlease snecify: | |
| Campus Status: | orcuse specify. | |
| Faculty Academic Professional/Staff Graduate | Student X Undergradu | ate Student |
| Visiting Scholar Other, please specify: | Stadent / Onder Brada | ate student |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid within last 3 years): 01/07/2021 | | |
| Additional training, <b>Date of Completion</b> (valid within last 5 years). 01/07/2021 | | |
| Role on Research Team (check all that apply): | | |
| Note on nesearch ream (check all that apply): | | |



## **Research Team**

| Recruiting Consenting Administering study pro | cedures 🔀 Hand | ling identifiable data |
|---|---|---|
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, etc | c.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | | |
| | <ul> <li>☑ This researcher is no longer an active research team member.</li> <li>Date added to research team: 07/26/2021 Date removed from research team: 05/06/2022</li> </ul> | |
| Date added to research team: 07/26/2021 Date | ate removed from | n research team: 05/06/2022 |
| Full Name: Margaret Danilovich | Degree: PhD | Dept. or Unit: |
| Professional Email: margaret.danilovich@cje.net | | hone: 217-300-5445 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign 🛛 Other, $\mu$ | olease specify: CJE | SeniorLife |
| Campus Status: | , | |
| Faculty Academic Professional/Staff Graduate | Student 🗌 Unde | rgraduate Student |
| ☐ Visiting Scholar ☐ Other, please specify: CJE SeniorLif | e Senior Director | of Research |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years): 9 | /13/2021 |
| Additional training, Date of Completion: | | |
| Role on Research Team (check all that apply): | | |
| Recruiting $igties$ Consenting $igties$ Administering study pro- | cedures 🔀 Hand | ling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, etc | c.), please specify the |
| procedure(s): | • | |
| This researcher should be copied on OPRS and IRB co | • | |
| This researcher is no longer an active research team | | |
| Date added to research team: 07/26/2021 | Date removed | from research team: |
| Full Name: Rachel Lessem | Degree: PhD | Dept. or Unit: |
| Professional Email: Rachel.Lessem@cje.net | | Dept. or Unit: hone: 773-508-1151 |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: | P | hone: 773-508-1151 |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, µ | P | hone: 773-508-1151 |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, µ Campus Status: | please specify: CJE | hone: 773-508-1151 SeniorLife |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate | Polease specify: CJE | hone: 773-508-1151 SeniorLife rgraduate Student |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLife | Polease specify: CJE | hone: 773-508-1151 SeniorLife rgraduate Student |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLif Training: | please specify: CJE<br>Student Unde<br>e Research and E | Hone: 773-508-1151 E SeniorLife Irgraduate Student valuation Associate |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLif Training: ☐ Required CITI Training, Date of Completion (valid with | please specify: CJE<br>Student Unde<br>e Research and E | Hone: 773-508-1151 E SeniorLife Irgraduate Student valuation Associate |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLift Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: | please specify: CJE<br>Student Unde<br>e Research and E | Hone: 773-508-1151 E SeniorLife Irgraduate Student valuation Associate |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, p. Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLift Training: ☒ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: Role on Research Team (check all that apply): | Polease specify: CJE Student Unde Research and E in last 3 years): 9 | Hone: 773-508-1151 E SeniorLife Irgraduate Student valuation Associate /13/2021 |
| Professional Email: Rachel.Lessem@cje.net Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☒ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate ☐ Visiting Scholar ☒ Other, please specify: CJE SeniorLif Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: | Polease specify: CJE Student Unde Research and E in last 3 years): 9 | Hone: 773-508-1151 E SeniorLife Irgraduate Student valuation Associate /13/2021 |



## **Research Team**

| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | | |
|---|---|---|---|
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB correspondence. | | | |
| This researcher is no longer an active research team member. | | | |
| Date added to research team: 07/26/2021 | Date added to research team: 07/26/2021 Date removed from research team: | | |
| Full Name: George Mois | <b>Degree:</b> PhD | | Dept. or Unit: |
| Professional Email: mois@illinois.edu | Degree in ind | Phone: 2 | 17-300-5445 |
| Campus Affiliation: | | | , 566 5115 |
| University of Illinois at Urbana-Champaign Other, p | lease specify: | | |
| Campus Status: | rease specify. | | |
| Faculty Academic Professional/Staff Graduate S | Student 🗆 Un | dergradua | ate Student |
| Visiting Scholar Other, please specify: CJE SeniorLife | | _ | |
| Training: | . researen ana | Lvaraatie | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | 02/05/20 | 120 |
| Additional training, <b>Date of Completion</b> : | iii iust s yeurs, | . 02, 03, 2 | ,20 |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study prod | edures 🕅 Hai | ndling ide | ntifiable data |
| Other, please specify: | eddies 🖂 Hai | iamig iac | Timable data |
| If administering biomedical study procedure (e.g., blood | draws scans | etc.). plea | se specify the |
| procedure(s): | araws, scaris, ( | cici,, pica | se speemy the |
| This researcher should be copied on OPRS and IRB co | rrespondence. | | |
| This researcher is no longer an active research team n | | | |
| Date added to research team: 08/31/2021 | | d from re | search team: |
| Full Name: Noah Olivero | Degree: | | Dept. or Unit: |
| | 2 08.00. | | |
| T Professional Fmail: noantoziwillinois.eou | | Phone: 2 | • |
| Professional Email: noahto2@illinois.edu Campus Affiliation: | | Phone: 2 | 17-300-5445 |
| Campus Affiliation: | lease specify: | Phone: 2 | • |
| Campus Affiliation: ☑ University of Illinois at Urbana-Champaign ☐ Other, p | lease specify: | Phone: 2 | • |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: | | | 17-300-5445 |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S | | | 17-300-5445 |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: | | | 17-300-5445 |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: | Student 🔀 Un | dergradua | 17-300-5445<br>ate Student |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: ☐ Required CITI Training, Date of Completion (valid with | Student 🔀 Un | dergradua | 17-300-5445<br>ate Student |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: | Student 🔀 Un | dergradua | 17-300-5445<br>ate Student |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: Role on Research Team (check all that apply): | Student 🔀 Un | dergradua<br>: 08/25/20 | 117-300-5445<br>ate Student |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: Role on Research Team (check all that apply): ☐ Recruiting ☐ Consenting ☒ Administering study processing ☐ Consenting ☒ Administering study processing ☐ Consenting ☐ Conse | Student 🔀 Un | dergradua<br>: 08/25/20 | 117-300-5445<br>ate Student |
| Campus Affiliation: ☐ University of Illinois at Urbana-Champaign ☐ Other, p Campus Status: ☐ Faculty ☐ Academic Professional/Staff ☐ Graduate S ☐ Visiting Scholar ☐ Other, please specify: Training: ☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion: Role on Research Team (check all that apply): | Student 🔀 Un | dergradua<br>: 08/25/20 | 117-300-5445<br>ate Student |

805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333-2670 irb@illinois.edu www.irb.illinois.edu Revised: 4/19/2021


| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | |
|---|---|---|
| procedure(s): This researcher should be copied on OPRS and IRB correspondence. | | |
| This researcher is no longer an active research team | | • |
| Date added to research team: 08/31/2021 | | ed from research team: |
| Date added to research team. 08/31/2021 | Date Telliov | eu iloili lesealcii tealii. |
| Full Names John Marandas | Dograda | Dont outlinit. |
| Full Name: John Marendes Professional Email: marendes@illinois.edu | Degree: | <b>Dept. or Unit: Phone:</b> 217-300-5445 |
| Campus Affiliation: | | Pnone: 217-300-3443 |
| ☐ University of Illinois at Urbana-Champaign ☐ Other, µ | nlease snecify: | |
| Campus Status: | neuse specify. | |
| Faculty Academic Professional/Staff Graduate | Student 🗆 Hn | dergraduate Student |
| Visiting Scholar Other, please specify: | | dergraduate Student |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 vears) | : 09/07/2021 |
| Additional training, <b>Date of Completion:</b> | , | , |
| Role on Research Team (check all that apply): | | |
| Recruiting Consenting Administering study pro | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | | · · |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | rrespondence | |
| This researcher is no longer an active research team | member. | |
| Date added to research team: 01/31/2022 | Date remove | ed from research team: |
| Full Name: Nithya Anand | Degree: | Dept. or Unit: |
| Professional Email: nithyas2@illinois.edu | • | Phone: 217-300-5445 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Other, µ | olease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate | Student 🔀 Un | dergraduate Student |
| ☐ Visiting Scholar ☐ Other, please specify: CJE SeniorLife Research and Evaluation Associate | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | : 08/25/2021 |
| Additional training, <b>Date of Completion:</b> | | |
| Role on Research Team (check all that apply): | <b>N</b> →7 | |
| igwedge Recruiting $igwidge$ Consenting $igwedge$ Administering study pro- | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | | |



### **Research Team**

| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | | |
|---|---|---|---|
| procedure(s): This researcher should be copied on OPRS and IRB correspondence. | | | |
| This researcher is no longer an active research team i | | d fuere u | esearch team: |
| Date added to research team: 01/31/2022 | Date remove | a from re | esearch team: |
| Full Names Vally Travillian | Dograda | | Dont author Applied |
| Full Name: Kelly Trevillian | Degree: | | <b>Dept. or Unit:</b> Applied Health Sciences- SHS |
| Professional Email: kellynt2@illinois.edu | | Phone: 1 | 217-265-6574 |
| Campus Affiliation: | | Phone: 2 | 217-203-0374 |
| ☐ University of Illinois at Urbana-Champaign ☐ Other, µ | ologco cnocify: | | |
| Campus Status: | neuse specify. | | |
| Faculty Academic Professional/Staff Graduate | Student M Una | deraradu | ata Student |
| Visiting Scholar Other, please specify: | ordaent 🖂 one | acigiada | ate student |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years): | 03/02/2 | 020 |
| Additional training, <b>Date of Completion</b> : | mi idat a yediaj. | 00,02,2 | 020 |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study pro- | cedures 🔀 Har | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, o | lepressio | n index, etc.), please |
| specify the procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | rrespondence. | | |
| This researcher is no longer an active research team I | | | |
| Date added to research team: 02/07/2022 D | ate removed fr | om resea | arch team: 05/06/2022 |
| Full Name: Alexandra Trekas | Degree: | | Dept. or Unit: Applied |
| | | | Health Sciences- SHS |
| Professional Email: trekas2@illinois.edu | | Phone: 2 | 217-265-6574 |
| Campus Affiliation: | | | |
| University of Illinois at Urbana-Champaign Urber, $\mu$ | olease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate Student Undergraduate Student | | | |
| ☐ Visiting Scholar ☐ Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, Date of Completion (valid with | in last 3 years): | 08/29/2 | 020 |
| Required CITI Training, <b>Date of Completion</b> (valid with Additional training, <b>Date of Completion</b> : | in last 3 years): | 08/29/2 | 020 |
| Required CITI Training, Date of Completion (valid with Additional training, Date of Completion: Role on Research Team (check all that apply): | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with Additional training, <b>Date of Completion</b> : | | | |

OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN

805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333-2670 irb@illinois.edu www.irb.illinois.edu Revised: 4/19/2021



### **Research Team**

| If administering biomedical study procedure (e.g., blood draws, scans, depression index, etc.), please | | |
|---|---|---|
| specify the procedure(s): | | |
| This researcher should be copied on OPRS and IRB correspondence. This researcher is no longer an active research team member. | | |
| Date added to research team: 02/07/2022 | | ed from research team: |
| Date added to research team. 02/07/2022 | Date lelliove | ed Holli research team. |
| Full Name: Vince Mathias | Dogradi | Dept. or Unit: |
| Professional Email: vmathias@illinois.edu | Degree: | Phone: 217-300-5445 |
| Campus Affiliation: | | Filone: 217-300-3443 |
| University of Illinois at Urbana-Champaign Other, | please specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate | Student Ur | ndergraduate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | nin last 3 years | ): 02/09/2022 |
| Additional training, Date of Completion: | | |
| Role on Research Team (check all that apply): | <u> </u> | |
| Recruiting Consenting Administering study pro | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB correspondence. This researcher is no longer an active research team member. | | |
| Date added to research team: 02/09/2022 Date removed from research team: | | |
| Date added to research team. 02/03/2022 | Date Telliov | ed from research team. |
| Full Name: Nathan Fensterheim | Degree: | Dept. or Unit: |
| Professional Email: nef4@illinois.edu | 208.00. | Phone: 217-300-5445 |
| Campus Affiliation: | | |
| ☐ University of Illinois at Urbana-Champaign ☐ Other, | please specify: | |
| Campus Status: | , | |
| Faculty Academic Professional/Staff Graduate | Student 🛛 Ur | ndergraduate Student |
| Visiting Scholar Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | nin last 3 years | ): 02/09/2022 |
| Additional training, Date of Completion: | | |
| Role on Research Team (check all that apply): | . 5 | |
| Recruiting Consenting Administering study pro | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | |
| procedure(s): | | |

OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN

805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333-2670 irb@illinois.edu www.irb.illinois.edu Revised: 4/19/2021



| This researcher should be copied on OPRS and IRB co | • | |
|---|---|---|
| This researcher is no longer an active research team | | |
| Date added to research team: 01/31/2022 | Date removed | from research team: 8/22/2022 |
| Full Name: Sharbel Yako | Degree: | Dept. or Unit: |
| Professional Email: syako2@illinois.edu | | <b>Phone:</b> 217-300-5445 |
| Campus Affiliation: | | |
| $\square$ University of Illinois at Urbana-Champaign $\square$ Other, $\mu$ | please specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate | Student 🔀 Un | dergraduate Student |
| Visiting Scholar Other, please specify: | | |
| Training: | | |
| ig Required CITI Training, <b>Date of Completion</b> (valid with | nin last 3 years) | : 02/09/2022 |
| Additional training, <b>Date of Completion:</b> | | |
| Role on Research Team (check all that apply): | | |
| ig Recruiting $igsquare$ Consenting $igsquare$ Administering study pro | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | rrespondence. | |
| This researcher is no longer an active research team | member. | |
| Date added to research team: 01/31/2022 | Date remove | ed from research team: |
| Full Name: Vinh Vo | Degree: | Dept. or Unit: |
| Professional Email: vinhvo2@illinois.edu | | Phone: 217-300-5445 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Other, | please specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate | Student 🔀 Un | dergraduate Student |
| Visiting Scholar Other, please specify: | _ | |
| Training: | | |
| Required CITI Training, Date of Completion (valid with | nin last 3 years) | : 10.22.2021 |
| Additional training, <b>Date of Completion</b> : | | |
| Role on Research Team (check all that apply): | | |
| Recruiting Consenting Administering study pro | cedures 🔀 Ha | ndling identifiable data |
| Other, please specify: | <del></del> | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), please specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | • | |
| This researcher is no longer an active research team | member. | |



### **Research Team**

Date added to research team: 05.20.2022 Date removed from research team: 8/22/2022

| | T | | T |
|---|---|---|---|
| Full Name: Zoe Faith Levitan | Degree: | Т | Dept. or Unit: |
| Professional Email: zfl2@illinois.edu | | Phone: 2 | 217-300-5445 |
| Campus Affiliation: | | | |
| $igert$ University of Illinois at Urbana-Champaign $igwdot$ Other, $\mu$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate | Student 🔀 Un | dergradua | ate Student |
| Visiting Scholar Other, please specify: | | | |
| Training: | | | |
| ig | in last 3 years) | : 05/13/2 | 022 |
| Additional training, Date of Completion: | | | |
| Role on Research Team (check all that apply): | | | |
| $ig igselow{igselow}$ Recruiting $igselow{igselow}$ Consenting $igotimes$ Administering study prod | cedures 🔀 Ha | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), plea | ise specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | • | | |
| This researcher is no longer an active research team r | nember. | | |
| Date added to research team: 05.20.2022 Date | removed from | research | team: |
| Full Name: Teresa Warren | Degree: BS | | Dept. or Unit: Applied |
| | | | Health Sciences- SHS |
| Professional Email: teresaw3@illinois.edu | | Phone: 2 | 217-265-6574 |
| Campus Affiliation: | | | |
| igert University of Illinois at Urbana-Champaign $igsqcup$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| 🔲 Faculty 🔲 Academic Professional/Staff 🔀 Graduate 🤉 | Student 🗌 Un | dergradua | ate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | | |
| Training: | | | |
| igwedge Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | : 06/02/2 | 022 |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| ig igotimes Recruiting $igotimes$ Consenting $igotimes$ Administering study prod | cedures 🔀 Ha | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), plea | se specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | rrespondence | | |



| This researcher is no longer an active research team r | nember. | | |
|---|---|---|---|
| Date added to research team: 06/15/2022 | Date remove | ed from re | esearch team: |
| Full Name: Summer Xia Yu | Degree: MSV | V | Dept. or Unit: Applied |
| | | | Health Sciences- SHS |
| Professional Email: xiayuyc2@illinois.edu | | Phone: 2 | 217-265-6574 |
| Campus Affiliation: | | | |
| igert University of Illinois at Urbana-Champaign $igsqcup$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff 🛛 Graduate S | Student 🔲 Un | dergradua | ate Student |
| Visiting Scholar Other, please specify: | | | |
| Training: | | | |
| $ig igselow{	extstyle igselow}{	ext{Required CITI Training, Date of Completion (valid with)}}$ | in last 3 years) | : 10/01/20 | 021 |
| Additional training, Date of Completion: | | | |
| Role on Research Team (check all that apply): | - | | |
| $ig igselow{igselow}{igselow}$ Recruiting $igotimes$ Consenting $igotimes$ Administering study prod | cedures 🔀 Ha | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), plea | se specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | • | 1 | |
| This researcher is no longer an active research team r | | | |
| Date added to research team: 06/15/2022 | Date remove | ed from re | esearch team: |
| | 1 | | |
| Full Name: Kori Trotter | Degree: BA | ı | Dept. or Unit: KCH |
| Professional Email: korit@illinois.edu | | Phone: 2 | 217-300-5445 |
| Campus Affiliation: | | | |
| igert University of Illinois at Urbana-Champaign $igwdot$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty 🛛 Academic Professional/Staff 🗌 Graduate S | Student 💹 Un | dergradua | ate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | : 4/25/22 | |
| Additional training, <b>Date of Completion</b> : | | | |
| Role on Research Team (check all that apply): | | | |
| ig igotimes Recruiting $igsqcup$ Consenting $igotimes$ Administering study prod | cedures 🔀 Ha | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), plea | se specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | • | • | |
| This researcher is no longer an active research team r | nember. | | |



| Date added to research team: 8/2/22 Da | te removed fro | m resear | ch team: |
|---|---|---|---|
| Full Name: Eliza Baby | Degree: MS | | Dept. or Unit: SHS |
| Professional Email: ebaby2@illinois.edu | | Phone: 2 | 17-265-6574 |
| Campus Affiliation: | | | |
| University of Illinois at Urbana-Champaign Other, I | please specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate | Student Un | dergradua | ite Student |
| Visiting Scholar Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | nin last 3 years) | : 08/21/20 | )22 |
| Additional training, Date of Completion: | | | |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study pro | cedures 🔀 Hai | ndling idei | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, | etc.), piea | se specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | • | | |
| This researcher is no longer an active research team | | | |
| Date added to research team: August 22, 2022 Date r | emovea from r | esearch t | eam: |
| Eull Namar Natalia Prana | Dogradi | | Dont or Unity CUC |
| Full Name: Natalia Rzepa Professional Email: nrzepa2@illinois.edu | Degree: | Phono: 3 | <b>Dept. or Unit:</b> SHS 17-265-6574 |
| Campus Affiliation: | | Filone. 2 | .17-203-0374 |
| University of Illinois at Urbana-Champaign Other, | nlease snecify: | | |
| Campus Status: | oicuse specijy. | | |
| II Faculty Academic Professional/Staff Graduate | Student Un | dergradua | ate Student |
| Faculty Academic Professional/Staff Graduate Visiting Scholar Other, please specify: | Student 🔀 Un | dergradua | ite Student |
| Visiting Scholar Other, please specify: | Student 🔀 Un | dergradua | ite Student |
| ☐ Visiting Scholar ☐ Other, please specify: Training: | | | |
| <ul> <li>□ Visiting Scholar □ Other, please specify:</li> <li>□ Training:</li> <li>□ Required CITI Training, Date of Completion (valid with</li> </ul> | | | |
| <ul> <li>□ Visiting Scholar □ Other, please specify:</li> <li>Training:</li> <li>□ Required CITI Training, Date of Completion (valid with □ Additional training, Date of Completion:</li> </ul> | | | |
| <ul> <li>□ Visiting Scholar □ Other, please specify:</li> <li>□ Training:</li> <li>□ Required CITI Training, Date of Completion (valid with</li> </ul> | nin last 3 years) | : Sept 13, | 2021 |
| <ul> <li>Visiting Scholar ☐ Other, please specify:</li> <li>Training:</li> <li>☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion:</li> <li>Role on Research Team (check all that apply):</li> </ul> | nin last 3 years) | : Sept 13, | 2021 |
| <ul> <li>Visiting Scholar ☐ Other, please specify:</li> <li>Training:</li> <li>☐ Required CITI Training, Date of Completion (valid with Additional training, Date of Completion:</li> <li>Role on Research Team (check all that apply):</li> <li>☐ Recruiting ☐ Consenting ☐ Administering study pro</li> </ul> | nin last 3 years)<br>cedures 🔀 Hal | : Sept 13, | 2021<br>ntifiable data |
| <ul> <li>Visiting Scholar ☐ Other, please specify:</li> <li>Training:</li> <li>☐ Required CITI Training, Date of Completion (valid with ☐ Additional training, Date of Completion:</li> <li>Role on Research Team (check all that apply):</li> <li>☐ Recruiting ☐ Consenting ☐ Administering study pro ☐ Other, please specify:</li> </ul> | nin last 3 years)<br>cedures 🔀 Hal | : Sept 13, | 2021<br>ntifiable data |
| <ul> <li>Visiting Scholar ☐ Other, please specify:</li> <li>Training:</li> <li>☐ Required CITI Training, Date of Completion (valid with Additional training, Date of Completion:</li> <li>Role on Research Team (check all that apply):</li> <li>☐ Recruiting ☐ Consenting ☐ Administering study pro Other, please specify:</li> <li>If administering biomedical study procedure (e.g., blood</li> </ul> | cedures Hal | : Sept 13,<br>ndling idel | 2021<br>ntifiable data |
| <ul> <li>Visiting Scholar ☐ Other, please specify:</li> <li>Training:</li> <li>☐ Required CITI Training, Date of Completion (valid with Additional training, Date of Completion:</li> <li>Role on Research Team (check all that apply):</li> <li>☐ Recruiting ☐ Consenting ☐ Administering study pro Other, please specify:</li> <li>If administering biomedical study procedure (e.g., blood procedure(s):</li> </ul> | nin last 3 years) cedures Hal | : Sept 13,<br>ndling idel | 2021<br>ntifiable data |



| Full Name: Ahmad Al-Juboory | Degree: | | Dept. or Unit: KCH |
|---|---|---|---|
| Professional Email: ahmada@illinois.edu | | Phone: 21 | 17-300-5445 |
| Campus Affiliation: | | | |
| University of Illinois at Urbana-Champaign Other, please specify: | | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Gradua | ate Student 🔀 U | ndergraduat | te Student |
| Visiting Scholar Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, Date of Completion (valid v | within last 3 years | ): August 26 | 5, 2022 |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| $\square$ Recruiting $\square$ Consenting $\square$ Administering study | procedures 🔀 Ha | andling iden | tifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blo | ood draws, scans | etc.), pleas | e specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRI | 3 correspondence | <b>:</b> . | |
| This researcher is no longer an active research tea | ım member. | | |
| Date added to research team: August 29, 2022 Da | te removed from | research te | am: |
| Full Name: James Shim | Degree: | | Dept. or Unit: SHS |
| Professional Email: jamesss3@illinois.edu | | Phone: | |
| Campus Affiliation: | | | |
| University of Illinois at Urbana-Champaign Other | er, please specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Gradua | ate Student 🔀 U | ndergraduat | te Student |
| Visiting Scholar Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, Date of Completion (valid v | within last 3 years | ): 08/31/22 | |
| Additional training, <b>Date of Completion</b> : | | | |
| Role on Research Team (check all that apply): | | | |
| Recruiting Consenting Administering study | procedures 🔀 Ha | andling iden | tifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blo | ood draws, scans | etc.), pleas | e specify the |
| procedure(s): | | | |
| This researcher should be copied on OPRS and IRI | 3 correspondence | ·. | |
| This researcher is no longer an active research tea | ım member. | | |
| Date added to research team: 9/9/22 | Date removed fr | om researcl | h team: |
| Full Name: Katie Naveja | Degree: | | Dept. or Unit: SHS |
| · | | | |
| OFFICE FOR THE PROTECTION OF RESEARCH SUBJECT | CTS UNIVERSITY OF ILLII | NOIS AT URBANA-C | HAMPAIGN |
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 T 217-333 | | | Revised: 4/19/2021 |



| Professional Email: knaveja2@illinois.edu | Phone | |
|---|---|---|
| Campus Affiliation: | | |
| $\square$ University of Illinois at Urbana-Champaign $\square$ Other, $p$ | lease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔀 Undergrad | uate Student |
| Visiting Scholar Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years): 8/28/2 | 2 |
| Additional training, <b>Date of Completion:</b> | | |
| Role on Research Team (check all that apply): | | |
| igert Recruiting $igwidge$ Consenting $igwedge$ Administering study proc | edures 🔀 Handling id | lentifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, etc.), ple | ease specify the |
| procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | • | |
| This researcher is no longer an active research team n | | |
| Date added to research team: 9/9/22 Date | e removed from resea | arch team: |
| Full Name: Afnaan Afsar Ali | Degree: | Dept. or Unit: |
| | | Department of |
| | | Kinesiology and |
| | | Community Health |
| Professional Email: aafsa2@illinois.edu | Phone | : 217-300-5445 |
| Campus Affiliation: | | |
| $\square$ University of Illinois at Urbana-Champaign $\square$ Other, $p$ | lease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔀 Undergrad | uate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | |
| Training: | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years): August | 21, 2022. |
| Additional training, <b>Date of Completion</b> : | | |
| Role on Research Team (check all that apply): | | |
| ig Recruiting $igsquare$ Consenting $igsquare$ Administering study proc | edures 🔀 Handling id | lentifiable data |
| Other, please specify: | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, depress | ion index, etc.), please |
| specify the procedure(s): | | |
| This researcher should be copied on OPRS and IRB co | • | |
| This researcher is no longer an active research team n | nember. | |
| Date added to research team: 10/12/2022 | Date removed from | m research team: |

| OFFICE FOR THE PROTECTION OF RESEAR | CH SUBJECTS | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 4/19/2021 |



| Full Name: Michael Varzino | Degree: | | Dept. or Unit: |
|---|---|---|---|
| | | | Department of |
| | | | Kinesiology and |
| | | | Community Health |
| Professional Email: varzino3@illinois.edu | | Phone: 2 | 17-300-5445 |
| Campus Affiliation: | | | |
| $\square$ University of Illinois at Urbana-Champaign $\square$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔀 Un | dergradua | ate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | | |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years): | Septemb | er 2, 2021 |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| igert oxtimes Recruiting $igwidge$ Consenting $igwedge$ Administering study prod | cedures 🔀 Har | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, o | depressio | n index, etc.), please |
| specify the procedure(s): | | | |
| This researcher should be copied on OPRS and IRB co | rrespondence. | | |
| This researcher is no longer an active research team r | nember. | | |
| Date added to research team: 10/12/2022 | Date remo | ved from | research team: |
| Full Name: Nila Silva de Albuquerque | <b>Degree:</b> PhD | | Dept. or Unit: |
| Professional Email: nila@illinois.edu | | Phone: 2 | 17-265-6574 |
| Campus Affiliation: | | | |
| $\square$ University of Illinois at Urbana-Champaign $\square$ Other, $p$ | lease specify: | | |
| Campus Status: | | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔲 Un | dergradua | ate Student |
| ☐ Visiting Scholar ☐ Other, please specify: Post-doctora | l research asso | ciate | |
| Training: | | | |
| Required CITI Training, <b>Date of Completion</b> (valid with | in last 3 years) | : 01/23/20 | 023 |
| Additional training, <b>Date of Completion:</b> | | | |
| Role on Research Team (check all that apply): | | | |
| ig Recruiting $ig $ Consenting $ig $ Administering study produced | cedures 🔀 Har | ndling ide | ntifiable data |
| Other, please specify: | | | |
| If administering biomedical study procedure (e.g., blood draws, scans, etc.), please specify the | | | |
| If administering biomedical study procedure (e.g., blood | draws, scans, o | etc.), plea | se specify the |
| procedure(s): | | | se specify the |
| procedure(s): This researcher should be copied on OPRS and IRB co | rrespondence. | | se specify the |
| procedure(s): | rrespondence. | | se specify the |



specify the procedure(s):

Date added to research team: 8/30/2022

### **Research Team**

Date removed from research team:

| Date added to research team: 01/28/2023 | Date removed from research team: | |
|---|---|---|
| Full Name: Maya Dye | Degree: | Dept. or Unit: |
| | | Department of |
| | | Kinesiology and |
| | | Community Health |
| Professional Email: mayadye2@illinois.edu | | <b>Phone:</b> 217-300-5445 |
| Campus Affiliation: | | |
| University of Illinois at Urbana-Champaign Other, p | lease specify: | |
| Campus Status: | | |
| Faculty Academic Professional/Staff Graduate S | Student 🔀 Un | dergraduate Student |
| ☐ Visiting Scholar ☐ Other, please specify: | | |
| Training: | | |
| Required CITI Training, Date of Completion (valid with | in last 3 years) | : August 21, 2023 |
| Additional training, <b>Date of Completion</b> : | | |
| Role on Research Team (check all that apply): | | |
| Recruiting Consenting Administering study prod | cedures 🔀 Hai | ndling identifiable data |
| Other places energy | | |

If administering biomedical study procedure (e.g., blood draws, scans, depression index, etc.), please

This researcher should be copied on OPRS and IRB correspondence.

This researcher is no longer an active research team member.

| OFFICE FOR THE PROTECTION OF RESEAR | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 4/19/202 |



For Engaging in a Collaborating Investigator Agreement for Individuals who are not Affiliated with an Institution that has an FWA

#### **COLLABORATOR INFORMATION**

| Collaborating Investigator's Name: Margaret Danilovich |
|-----------------------------------------------------------|
| Collaborating Investigator's Institution (if applicable): |
| CITI Training Completion Date: Sept 13, 2021 |

#### PROTOCOL INFORMATION

| The above is a Collaborating Investigator in the following research study being conducted by the University |
|---|
| of Illinois at Urbana-Champaign: |
| Illinois Principal Investigator: Dr. Wendy Rogers |
| Illinois Protocol Number: 22212 |
| Illinois Title: Video Technology-based Social Engagement |
| Illinois PI Home Unit (DMI Unit Name): Applied Health Sciences |

I acknowledge and agree that the University of Illinois at Urbana-Champaign Principal Investigator will direct and supervise my research activities outside the Illinois campus.

I have reviewed the following documents: (a) The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, available at <a href="http://ohsr.od.nih.gov/guidelines/belmont.html">http://ohsr.od.nih.gov/guidelines/belmont.html</a>; (b) the U.S. Department of Health and Human Services (HHS) regulations for the Protection of Human Subjects at 45 CFR part 46; and (c) the terms of Illinois's FWA; and (d) the Illinois policies and procedures for the protection of human subjects, available at <a href="https://oprs.research.illinois.edu/">https://oprs.research.illinois.edu/</a>. I understand and accept my responsibility to comply with the standards and requirements set forth in the above-identified documents and to protect the rights and welfare of human subjects involved in the Research.

I will comply with all applicable international, federal, state, and local laws, regulations and policies that may provide additional protection for human subjects participating in the Research.

I will abide by all determinations of the Illinois Institutional Review Board (IRB) and will accept the final authority and decisions of the IRB, including but not limited to directives to terminate participation in the Research.

I will complete any educational training required by Illinois and the IRB prior to initiating activities related to the Research.

I will not enroll subjects in the Research prior to its review and approval by the IRB.

| OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS | | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 11/11/2019 |



I will report promptly to the IRB any proposed changes in the Research. I will not initiate changes in the Research without prior IRB review and approval, except where necessary to eliminate apparent immediate hazards to subjects.

When responsible for enrolling subjects, I will obtain, document and maintain records of informed consent for each such subject or each subject's legally authorized representative as required by HHS regulations at 45 CFR part 46 and as described in the Research protocol approved by the IRB.

I will report immediately to the IRB any unanticipated problems involving risks to subjects or others in the Research.

I acknowledge the IRB's responsibility for initial and continuing review, recordkeeping, reporting, and certification for the Research. I will cooperate fully with the IRB and will provide all information requested by the IRB in a timely fashion.

I acknowledge my responsibility for safeguarding the rights and welfare of each Research subject and that the subject's rights and welfare must take precedence over the goals and requirements of the Research.

| Collaborating | Individual Investigator's Signatur | e: | Many | Pul | Date: 8.30.21 |
|---|---|---|---|---|---|
| | : <u>Margaret Danilovich</u> Degrees: <u>DP</u><br>: <u>Margaret.danilovich@cje.net</u> | T, PhD | | | |
| Institution is a | Investigator's Institution (if appli<br>uthorized to conduct the Research | n at this Inst | titution und | er the terms of | |
| Authorized In:<br>Printed Name<br>Complete Add | | | | | |
| For Illinois:<br>Illinois PI Dep | artment Head<br>Yum' C. Arabes | | | | |
| Signature: | | | | Date: | 08/31/2021` |
| | : Kim C. Graber<br>Kinesiology and Community Hea | lth | | | |
| _ | OFFICE FOR THE PROTECTION OF RESEAS | RCH SUBJECTS | UNIVERSITY OF IL | LINOIS AT URBANA-CHA | |
| 80 | 05 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu Re | vised: 11/11/2019 |



\*If signing as a delegate, please include name and title below: Name:

Title:

Office of the Vice Chancellor for Research

Susan A. Martinis, Ph.D; Vice Chancellor for Research Office of Vice Chancellor for Research 601 E John Street Champaign, IL 61820



irb@illinois.edu



For Engaging in a Collaborating Investigator Agreement for Individuals who are not Affiliated with an Institution that has an FWA

#### **COLLABORATOR INFORMATION**

| Collaborating Investigator's Name: | Rachel Lessem | |
|------------------------------------------|------------------|----------------|
| Collaborating Investigator's Institution | (if applicable): | CJE SeniorLife |
| CITI Training Completion Date: Sept 13, | 2021 | |

#### PROTOCOL INFORMATION

| The above is a Collaborating Investigator in the following research study being conducted by the University |
|---|
| of Illinois at Urbana-Champaign: |
| Illinois Principal Investigator: Dr. Wendy Rogers |
| Illinois Protocol Number: 22212 |
| Illinois Title: Video Technology-based Social Engagement |
| Illinois PI Home Unit (DMI Unit Name): Applied Health Sciences |

I acknowledge and agree that the University of Illinois at Urbana-Champaign Principal Investigator will direct and supervise my research activities outside the Illinois campus.

I have reviewed the following documents: (a) The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, available at <a href="http://ohsr.od.nih.gov/guidelines/belmont.html">http://ohsr.od.nih.gov/guidelines/belmont.html</a>; (b) the U.S. Department of Health and Human Services (HHS) regulations for the Protection of Human Subjects at 45 CFR part 46; and (c) the terms of Illinois's FWA; and (d) the Illinois policies and procedures for the protection of human subjects, available at <a href="https://oprs.research.illinois.edu/">https://oprs.research.illinois.edu/</a>. I understand and accept my responsibility to comply with the standards and requirements set forth in the above-identified documents and to protect the rights and welfare of human subjects involved in the Research.

I will comply with all applicable international, federal, state, and local laws, regulations and policies that may provide additional protection for human subjects participating in the Research.

I will abide by all determinations of the Illinois Institutional Review Board (IRB) and will accept the final authority and decisions of the IRB, including but not limited to directives to terminate participation in the Research.

I will complete any educational training required by Illinois and the IRB prior to initiating activities related to the Research.

I will not enroll subjects in the Research prior to its review and approval by the IRB.

| OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS | | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 11/11/2019 |



I will report promptly to the IRB any proposed changes in the Research. I will not initiate changes in the Research without prior IRB review and approval, except where necessary to eliminate apparent immediate hazards to subjects.

When responsible for enrolling subjects, I will obtain, document and maintain records of informed consent for each such subject or each subject's legally authorized representative as required by HHS regulations at 45 CFR part 46 and as described in the Research protocol approved by the IRB.

I will report immediately to the IRB any unanticipated problems involving risks to subjects or others in the Research.

I acknowledge the IRB's responsibility for initial and continuing review, recordkeeping, reporting, and certification for the Research. I will cooperate fully with the IRB and will provide all information requested by the IRB in a timely fashion.

I acknowledge my responsibility for safeguarding the rights and welfare of each Research subject and that the subject's rights and welfare must take precedence over the goals and requirements of the Research.

| | · | | • | • | | |
|---|---|---|---|---|---|---|
| Collaborating I | ndividual Investigator's Signatur | e: | Parkelo | Tessin | _ Date: | 8/30/2021 |
| | Rachel N. Lessem Degrees: JD, Ph<br>Rachel.Lessem@cje.net | <u>ıD</u> | | | | |
| | nvestigator's Institution (if application) application (if application) application (if application) are set of the second conduct the Research (in the second conduct the Research (in the second conduct the Research (in the second conduct the Research (in the second conduct the Research (in the second conduct the second conduct the Research (in the second conduct the seco | | | | | |
| Kum | C. Kraber | | | | | |
| Ву:/ | | | | [ | Date: <u>08/3</u> | 31/2021 |
| Authorized Ins | titutional Signatory | | | | | |
| Printed Name: | <u>Kim C. Graber</u> | | | | | |
| Complete Addr | ress: Kinesiology and Community | <u>Health</u> | | | | |
| For Illinois: | | | | | | |
| Illinois PI Depa | rtment Head | | | | | |
| Signature: | | Da | te: | | | |
| Printed Name: | | | | | | |
| Department: | | | | | | |
| *If signing as a | delegate, please include name ar | nd title belo | w: | | | |
| Name: | | | | | | |
| _ | OFFICE FOR THE PROTECTION OF RESEAR | RCH SUBJECTS | UNIVERSITY OF IL | LINOIS AT URBANA | A-CHAMPAIGN | |
| 905 | West Pennsylvania Avenue MC 005 Urbana II 61901 | T 247 222 2670 | ich Cillingia adu | varavida illinaia ada | Revised: 11 | /11/2010 |



Title:

#### Office of the Vice Chancellor for Research

Susan A. Martinis, Ph.D; Vice Chancellor for Research Office of Vice Chancellor for Research 601 E John Street Champaign, IL 61820





#### **Letter of Agreement for Senior Housing Communities**

| I,Margaret Danilovich_ (print your name), of <u>CJE Senic</u> grant permission to researchers from the Aging and Neurocogn and Aging Lab at the University of Illinois Urbana-Champaign to collect data at CJE SeniorLife facilities. | ition Lab and Human Factors |
|---|---|
| This agreement will be in effect through August 2024. | |
| Margaret Danilovich<br>Printed name | _ |
| Marthal | 8.4.21 |
| Signature | Date |
| Please return this letter to Dr. Raksha Mudar via: | |

Email: raksha@illinois.edu

Address: 901 S Sixth St Champaign, IL 61820

Please call Raksha Mudar (217-333-4718) if you have any questions about this form and/or study.